# **Statistical Analysis Plan**

# A PHASE II, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, MULTICENTER STUDY TO ASSESS THE SAFETY AND EFFICACY OF VM202 IN SUBJECTS WITH CRITICAL LIMB ISCHEMIA

Protocol VMCLI-II-09-002 July 28, 2011

| Sponsor: | |
|--------------|------------------|
| Prepared by: | |
| Varsion | October 2nd 2013 |

# TABLE OF CONTENTS

| LIS | ST OF ABBREVIATIONS | 4 |
|---|---|---|
| DE | FINITIONS | 6 |
| 1. | INTRODUCTION | 7 |
| 2. | OBJECTIVES | 7 |
| | 2.1. Primary Objective | |
| | 2.2. SECONDARY OBJECTIVES | |
| 3. | STUDY OVERVIEW | 7 |
| 4. | SAMPLE SIZE JUSTIFICATION | 10 |
| 5. | GENERAL ANALYSIS CONSIDERATIONS | 10 |
| | 5.1. VISIT WINDOWS | 10 |
| | 5.2. STATISTICAL METHODS | |
| | 5.3. UNMASKING OF THE RANDOMIZATION CODES | |
| 6. | ANALYSIS POPULATIONS | 11 |
| 7. | SUBJECT DISPOSITION | 12 |
| 8. | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 12 |
| 9. | MEDICAL HISTORY | 13 |
| 10. | EFFICACY ANALYSES | 13 |
| | 10.1. Primary Efficacy Variable | |
| | 10.1.1. Subgroup Analysis | |
| | 10.1.2. Imputation Methods of VAS Results for the ITT Population | 14 |
| | 10.2. SECONDARY EFFICACY VARIABLES | |
| | 10.2.1. VISUAL ANALOGUE SCALE FOR PAIN (VAS) | |
| | 10.2.2. TRANSCUTANEOUS OXYGEN PRESSURE ASSESSMENT (TCPO <sub>2</sub> , MMHg) | |
| | 10.2.3. HEMODYNAMIC ASSESSMENTS (ABI/TBI) | |
| | 10.2.5. WOUND HEALING AND ULCER MEASUREMENT | |
| | 10.2.6. QUALITY OF LIFE (VASCUQOL) | |
| | 10.2.7. Amputation and Mortality Rate | |
| | 10.2.8. Rutherford Classification | |
| | 10.3. BASELINE VALUES | |
| | 10.4. MULTIPLICITY ADJUSTMENTS | _ |
| 11. | SAFETY ANALYSES | |
| | 11.1. STUDY DRUG EXPOSURE | _ |
| | 11.2. ADVERSE EVENTS | |
| | 11.4. VITAL SIGNS | |
| | 11.5. RETINAL FUNDOSCOPY | |

| 11.6. INJECTION SITE REACTION | 24 |
|-----------------------------------------|----|
| 11.6. INJECTION SITE REACTION | |
| 11.8. Interim Analyses | 26 |
| APPENDIX A: LIST OF TABLES AND LISTINGS | 27 |
| APPENDIX B: TABLE LAYOUTS | 33 |
| APPENDIX C: FIGURE LAYOUTS | 69 |
| APPENDIX D: LISTING LAYOUTS | 71 |

#### LIST OF ABBREVIATIONS

ABI ankle-brachial index

AE adverse event

ALT alanine transaminase (SGPT)

ANOVA analysis of variance

AST aspartate transaminase (SGOT)

BP blood pressure
BUN blood urea nitrogen
CBC complete blood count
CI confidence interval
CLI critical limb ischemia

cm centimeter(s)

CSR clinical study report CRF case report form DNA deoxyribonucleic acid

D day(s)

DSMB Data Safety Monitoring Board HGF hepatocyte growth factor

IM intra-muscular ITT intent-to-treat

IRB Institutional Review Board LSD least significant difference

MedDra Medical Dictionary for Regulatory Activities

mg Milligrams

mmHg milligrams of mercury

MRA magnetic resonance angiography

 $\begin{array}{ll} N & \quad & \text{Number} \\ \text{Ng} & \quad & \text{nanogram(s)} \\ \text{O}_2 & \quad & \text{Oxygen} \end{array}$ 

PAD peripheral artery disease pH hydrogen ion concentration

PP per-protocol

PTA percutaneous transluminal angioplasty

RBC red blood count
SAE serious adverse event
SAP Statistical Analysis Plan

sDBP sitting diastolic blood pressure

SGPT serum glutamic pyruvic transaminase (same as ALT)

# LIST OF ABBREVIATIONS (CONTINUED)

SOC System Organ Class

SVR systemic vascular resistance

TBI toe-brachial index

TcPO<sub>2</sub> Transcutaneous Oxygen Pressure Assessment

VAS visual analog scale

VEGF vascular endothelial growth factor

vs. Versus

WBC white blood count WFI water for injection

#### **DEFINITIONS**

Adverse Event An adverse event (AE) is the development of an undesirable

medical condition following or during exposure to a pharmaceutical product, whether or not it is considered

causally related to the product.

Baseline The last non-missing value prior to first dose of study drug. Serious AE An AE occurring at any dose that: results in death; is a

An AE occurring at any dose that: results in death; is a life-threatening experience; requires hospitalization or prolongation of an existing hospitalization; results in a persistent or significant disability/incapacity; or is a

congenital anomaly/birth defect in the offspring of a subject

who received study drug.

Treatment-emergent AE AEs with an onset time after the initial dose of study drug.

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of VM BioPharma Protocol VMCLI-II-09-002 [A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multi-center Study to Assess the Safety and Efficacy of VM202 in Subjects with Critical Limb Ischemia]. The purpose of this plan is to provide specific guidelines from which the analysis will proceed. Any deviations from these guidelines will be documented in the clinical study report (CSR).

#### 2. OBJECTIVES

## 2.1. Primary Objective

The primary objective of this analysis is to evaluate the safety of IM administration of VM202 in subjects with moderate or high-risk CLI (Rutherford Clinical Severity Score equal to 4 or 5) who are poor or non-candidates for surgical or percutaneous revascularization.

## 2.2. Secondary Objectives

The secondary objective of the study is to evaluate potential bioactivity of IM administration of VM202 in subjects with CLI, when compared to placebo, on:

- Change in VAS for pain at rest
- Leg ulcer healing (as assessed by ulcer surface area and time to complete healing)
- Hemodynamic assessment (ABI/TBI)
- Tissue oxygenation (TcPO<sub>2</sub>)
- Incidence and extent of lower leg amputation, limb salvage or other surgical interventions
- VascuQoL
- Perfusion (MRA)

#### 3. STUDY OVERVIEW

This is a 12 month Phase II, double-blind, randomized, placebo-controlled, multi-center study designed to assess the safety and efficacy of VM202 in subjects with critical limb ischemia.

Subjects who meet the eligibility criteria will be randomized in a 2:2:1 ratio to one of three treatment arms: Low Dose (8 mg VM202), High Dose (16 mg VM202) or placebo, respectively.

Subjects in the Low Dose Group (8 mg VM202) will receive:

- Day 0: 4 mg of VM202 (16 injections of 0.5 ml of VM202)
- Day 14: 4 mg of VM202 (16 injections of 0.5 ml of VM202)
- Day 28: Placebo only (16 injection of 0.5 ml normal saline)
- Day 42: Placebo only (16 injection of 0.5 ml normal saline)

Subjects in the High Dose Group (16 mg VM202) will receive:

- Day 0: 4 mg of VM202 (16 injections of 0.5 ml of VM202)
- Day 14: 4 mg of VM202 (16 injections of 0.5 ml of VM202)
- Day 28: 4 mg of VM202 (16 injections of 0.5 ml of VM202)
- Day 42: 4 mg of VM202 (16 injections of 0.5 ml of VM202)

Subjects in the placebo control group will receive 16 injections of 0.5 ml normal saline at each visit.

Table 1 lists the final dose and dose per visit to be administered by study arm.

Table 1. VM202 administration for each study arm

| TREATMENT | FINAL DOSE | Do | OSE VM202 | (MG) PER V | ISIT |
|---|---|---|---|---|---|
| GROUP | VM202 | DAY 0 | <b>DAY 14</b> | <b>DAY 28</b> | <b>DAY 42</b> |
| Low Dose | 8 mg | 4 | 4 | 0 | 0 |
| High Dose | 16 mg | 4 | 4 | 4 | 4 |
| Placebo | 0 | 0 | 0 | 0 | 0 |

The schedule of study visits and the clinical parameters that will be measured at the visits are summarized in Table 2 below.

TABLE 2 SCHEDULE OF EVALUATIONS AND VISITS

| Procedure | Screening /<br>Baseline | 1 <sup>st</sup> Inj<br>Da | ection<br>y 0 | 2 <sup>nd</sup> In<br>Day 1 | jection<br>4 ± 3 D | 3 <sup>rd</sup> Inj<br>Day 28 | ection<br>8 ± 3 D | 4 <sup>th</sup> Inj<br>Day 42 | jection<br>2 ± 3 D | <b>Day 49</b> | <b>Day 90</b> | 6 mo | 9 mo | 12 mo | Early |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| FROCEDURE | (-30 – 0 D) | Pre-<br>dose | Post-<br>dose | Pre-<br>dose | Post-<br>dose | Pre-<br>dose | Post-<br>dose | Pre-<br>dose | Post-<br>dose | ± 3 D | ± 7 D | ± 1 mo | ± 1 mo | ± 1 mo | Withdrawal |
| <b>Baseline Evaluation</b> | | | | | | | | | | | | | | | |
| Informed Consent | ✓ | | | | | | | | | | | | | | |
| Complete Medical History | ✓ | | | | | | | | | | | | | | |
| Complete Physical Exam | ✓ | | | | | | | | | | | | | | |
| Cancer screening <sup>†</sup> | ✓ | | | | | | | | | | | | | | |
| Viral screening – HIV, HTLV, HBV, HCV | <b>✓</b> | | | | | | | | | | | | | | |
| Urinalysis | ✓ | | | | | | | | | | | | | | |
| ECG | ✓ | | | | | | | | | | | | | | |
| Pregnancy test | ✓ | | | | | | | | | | | | | | |
| Safety and Efficacy Parameters | | | | | | | | | | | | | | | |
| Retinal Fundoscopy | ✓ | | | | | | | | | | | | | ✓ | ✓ |
| Vital Signs | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Concomitant Medications | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | ✓ | ✓ | <b>✓</b> | ✓ | ✓ |
| Serum Chemistry and hematology | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | ✓ | ✓ | <b>√</b> | ✓ | ✓ |
| Photograph and measurement of ulcer(s) <sup>††</sup> | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Visual Analog Scale (VAS) score | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | | ✓ | ✓ | ✓ | ✓ | |
| ABI/TBI | ✓ | ✓ | | | | ✓ | | | | | ✓ | ✓ | ✓ | ✓ | |
| TcPO <sub>2</sub> | ✓ | ✓ | | | | | | | | | | ✓ | <b>✓</b> | ✓ | |
| VascuQol | | ✓ | | | | | | | | | ✓ | | <b>✓</b> | ✓ | |
| Copies of VM202 in whole blood | | ✓ | <b>√</b> ** | | | | | ✓ | <b>√</b> ** | ✓ | ✓ | ✓ | | | <b>√</b> ¹ |
| Rutherford Classification | ✓ | | | | | | | | | | | ✓ | ✓ | ✓ | |
| Serum HGF | | ✓ | | | | | | ✓ | | ✓ | ✓ | | | | <b>√</b> ¹ |
| MRA (at designated site(s) only) | | ✓ | | | | | | | | | | ✓ | ✓ | | |
| Treatment | | | | | | | | | | | | | | | |
| Injection site reaction assessment | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | | | | <b>√</b> <sup>2</sup> |
| Adverse Events | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |

<sup>†</sup> Includes: cancer markers (carcinoembryonic antigen (CEA), alpha fetoprotein (AFP), CA19-9, and CA125 (females only)); chest X-ray or CT scan of the chest (if subject has a previous history of tobacco use, a CT scan will be performed instead of the chest X-ray) within 3 months; pap smear and mammogram if not performed within past 12 months (females only); PSA (males only); for subjects  $\geq$  50 years old, colonoscopy within past 10 years

<sup>††</sup> If present prior to first study drug administration

<sup>\*\* 2</sup> hours after injection (± 1 hour)

<sup>1</sup> If withdrawal occurred before Day 90 Visit

<sup>2</sup> If withdrawal occurred before Day 49 Visit

## 4. SAMPLE SIZE JUSTIFICATION

The sample size for this Phase 2 study was chosen to estimate effect sizes and variability for a pivotal study. Assuming a standard deviation for change in VAS scores of 25, a mean change of 30 in the high dose group, 28 in the low dose group, and 10 in the placebo group, an Analysis of Variance (ANOVA) F-test at alpha of 5%, a sample size of 20:20:10 for high dose, low dose and placebo, respectively, will have 49% power to detect an overall difference among treatment groups.

## 5. GENERAL ANALYSIS CONSIDERATIONS

The statistical analyses will be reported using summary tables, figures, and data listings. Continuous variables will be summarized with means, standard deviations, standard error, medians, minimums, and maximums for each treatment arm. Categorical variables will be summarized by counts and by percentage of subjects in corresponding categories.

All analyses and tabulations will be performed using SAS<sup>®</sup> Version 9.1 or higher on a PC platform. Tables and listings will be presented in RTF format.

#### 5.1. Visit Windows

Data at each scheduled follow up visit will be analyzed according to the nominal visit identified on the CRF, regardless of the actual elapsed time since treatment.

#### 5.2. Statistical Methods

Two-sided p-values < 0.05 will be considered statistically significant, unless otherwise stated.

Separate statistical tests will be performed at each time point for key endpoints of interest.

In general, an overall test to determine if there is a statistically significant difference among the three treatment arms will be conducted first. Further comparisons will be made to determine if either the low or high dose groups are significantly different from the placebo group.

For continuous variables, a one-way analysis of variance (ANOVA) with treatment group (high dose, low dose, and placebo) as a factor will be used to determine if there is a significant difference among the groups. The low and high dose groups will each be compared against the placebo group using Dunnett's test. The mean difference between the VM202 groups versus placebo along with 95% confidence intervals for the mean difference will also be presented. To be viewed as secondary, an additional set of analyses will be run using non-parametric tests. A Jonckheere-Tepstra test will be applied to the VAS change from baseline results to detect overall trend differences. Non-parametric pairwise treatment comparisons versus placebo will also be made using Wilcoxon Rank Sum test. Within each treatment group for each endpoint, both a paired t-test (parametric) and Wilcoxon Signed Rank test will be run to test for differences comparing baseline to each post-baseline assessment.

For categorical variables, Fisher's exact test will be used to determine if there is a significant difference among the three treatment groups. Separate Fisher's exact tests will be used to compare the low and high dose groups to the placebo group.

For time-to-event variables (such as amputation, limb salvage and mortality), Kaplan-Meier estimates will be used to estimate survival times. Differences in survival times will be compared among groups using the log-rank test.

## 5.3. Unmasking of the Randomization Codes

The complete randomization code will be unmasked after all the data queries related to the efficacy and safety outcomes have been resolved and the corresponding data revisions have been completed in the database. The DSMB Chair will review a limited set of unblinded tables and listings through DSMB meetings. The analyses for the DSMB meeting will be performed by an independent clinical research organization

## 6. ANALYSIS POPULATIONS

The following subject populations will be used for analysis:

The Intent-to-Treat (ITT) population will include all subjects who were randomized regardless of whether treatment was received. Subjects will be analyzed according to the treatment to which they were randomized.

The Safety population will include all subjects who receive at least one dose of study drug medication and data will be analyzed according to the treatment actually received. The safety analyses will be performed on the Safety population.

The per-protocol (PP) population will include all subjects who received the correct dose of study drug medication, have the 9-month VAS assessment, and do not have any protocol violations or major deviations as determined by Medical Monitoring. The per-protocol population will be determined in a blinded review before database lock. Subjects will be analyzed according to the treatment to which they were randomized. Primary efficacy analyses will be performed on the PP population.

## 7. SUBJECT DISPOSITION

Subject disposition information will be summarized for all subjects by dose cohort. Summaries will include the number of subjects:

- enrolled (overall)
- in each analysis population
- who received all planned doses of VM202
- last visit attended (Note: subject considered to have attended a visit if at least one assessment was reported for that visit)
- who completed the study (as determined by Study Exit Status page)
- primary reason for discontinuation for those who did not complete the study

## 8. DEMOGRAPHIC AND BASELINE CHARACTERISTICS

Demographic and baseline characteristics will be summarized for the ITT, Safety and PP analysis populations. Demographic variables include:

- age at informed consent
- sex
- race

Baseline variables will include height, weight, and incidence of diabetes mellitus and renal dysfunction. Age, height and weight will be compared among treatment groups (overall

comparison) using the method for continuous variables. All other variables will be compared among groups (overall comparison) using the method for categorical variables.

## 9. MEDICAL HISTORY

Medical history will be categorized by body system. Medical history and peripheral vascular disease intervention history at baseline will be summarized by frequencies and rates on the Safety population.

## 10. EFFICACY ANALYSES

The primary efficacy analysis will be based on the PP analysis population. Additional efficacy analyses will be performed on the ITT population.

## 10.1. Primary Efficacy Variable

Subjects will be asked to assess the level of pain they feel by placing a perpendicular line on a scale of 0 (No Pain) to 100 (Pain as bad as it can be) at each visit. The subject's Visual Analogue Scale (VAS) score will be determined by where the subject places the perpendicular line by two independent readers. The average scores from the two readers will be used as the pain score for the corresponding subject. If a score is reported by only one reader, then that score will be assigned as the pain score. The primary efficacy endpoint is the change in pain level between baseline and the 9-month follow-up as determined by VAS. The change in pain will be calculated for each subject as follows:

Change = 
$$9$$
-month VAS – Baseline VAS

Since higher VAS indicates worse pain, a negative value of change means an improvement, and a positive value of change means deterioration.

The mean change in pain will be compared among the three treatment groups. The statistical null and alternative hypotheses for the primary efficacy endpoint are:

$$H_o$$
:  $\mu_H = \mu_L = \mu_P$  and  $H_a$ : at least one of the three  $\mu$ 's is different,

where  $\mu_H$ ,  $\mu_L$ , and  $\mu_P$  are mean change in pain from baseline to 9-month follow-up for VM202 high dose, VM202 low dose, and placebo groups, respectively.

One-way Analysis of Variance (ANOVA) with treatment (VM202 high dose, VM202 low dose, and placebo) as the factor will be used to compare the mean change in pain among the three treatment groups. Dunnett's test will be used to compare the mean change in pain level between VM202 high dose to placebo and between VM202 low dose to placebo. This analysis will be repeated using Percent (%) Change from Baseline, where Percent Change from Baseline is defined as:

• % Change from Baseline = [ (9 month VAS – Baseline VAS)/Baseline VAS]\* 100

An additional set of analyses will be run using non-parametric tests as described in Section 5.2 for continuous variables.

## 10.1.1. Subgroup Analysis

It is clinically considered that sex and co-morbidities (diabetes or renal dysfunction) can affect the change in pain. A two-factor ANOVA with treatment and one of the covariates (sex, diabetes, or renal dysfunction) as the factors will be used to analyze the primary endpoint. For each analysis, treatment group, covariate, and treatment group by covariate interaction will be included in the model. If the treatment by covariate interaction is judged to be insignificant (p > 0.10) then the interaction term will be removed from the model and pairwise treatment comparisons of adjusted means vs. Placebo using Dunnett's test will be presented. If the treatment by covariate interaction term is significant, then separate analyses will be performed for the different levels of the covariate of consideration.

## 10.1.2. Imputation Methods of VAS Results for the ITT Population

In order to include all subjects in the ITT population, the following imputation rules will be applied for analysis of the ITT population.

For subjects without the primary efficacy endpoint (VAS change from baseline to 9 months), the following imputation methods will be applied:

- For missing Baseline VAS, assign the VAS score at Screening if the VAS score at Day 0 is missing.
- For missing 9 month VAS, assign the 12 month VAS score if the 9 month VAS is missing.

• For missing 9 month VAS, assign the last reported VAS prior to the 9 month VAS visit if both the 9 month and 12 month VAS assessments are missing.

For subjects who had a major amputation or limb procedure carried out, the following imputation methods will be applied:

- For subjects with a major amputation, assign the post baseline VAS score prior to the amputation.
- For subjects with a limb salvage, assign the post baseline VAS score prior to the intervention.

## 10.2. Secondary Efficacy Variables

The analyses for the secondary efficacy variables will be performed based on the Per-Protocol Population and ITT Populations. The secondary efficacy endpoints include:

## 10.2.1. VISUAL ANALOGUE SCALE FOR PAIN (VAS)

The VAS measurements, change from baseline and percent change from baseline will be summarized at each visit by treatment arm using the methods described in Section 10.1.

Categorical analysis of VAS measurements will be performed by visit. Each VAS measurement will be assigned to one of the following 4 categories: 0-4 mm, 5-44 mm, 45-74 mm and 75-100 mm. Incidence and percentage of each VAS category will be presented for Baseline and each post baseline visit. Testing for treatment differences versus placebo will be carried out using a CMH test (Row Means Score).

## 10.2.1.1 Imputation Methods of VAS Results for the ITT Population

For subjects without the efficacy endpoint (VAS change from baseline to any post baseline result), the following imputation methods will be applied:

- For missing Baseline VAS, assign the VAS score at Screening if the VAS score at Day 0 is missing.
- For any post baseline VAS, assign the post baseline VAS score prior to the missing post baseline VAS via the last observation carried forward (LOCF) method.

For subjects who had a major amputation or limb procedure carried out, the following imputation methods will be applied:

- For subjects with a major amputation, assign the VAS score prior to the amputation.
- For subjects with a limb salvage, assign the VAS score prior to the intervention.

## 10.2.2. Transcutaneous Oxygen Pressure Assessment (TcPO<sub>2</sub>, mmHg)

Transcutaneous oxygen pressure measurements (tissue oxygenation) will be measured at the anterior calf, posterior calf, dorsum foot and chest.  $TcPO_2$  measurements and change from baseline (= post-treatment – baseline) for each body region will be summarized by study visit and treatment arm using the method for continuous variables. The baseline value is the measurement taken at the Day 0 (Pre-Dose) Visit if the percent difference (=|Day 0 – Screening|/Screening×100%) between the measurements taken at the Screening Visit and the Day 0 Visit is  $\leq 15\%$ . Otherwise, the baseline value is the average of the measurements taken at Screening and Day 0 Visits.

Additionally, TcPO<sub>2</sub> ratio for each of the body region (anterior calf, posterior calf, and dorsum foot) to chest will be calculated for each subject as TcPO<sub>2</sub> at each body region divided by the TcPO<sub>2</sub> at chest. The chest value to be used as the denominator when generating the TcPO<sub>2</sub> ratio for each of the body region will be by subject and calculated by taking the average of that subject's non-missing chest results reported at Day 0, Day 180, Day 270 and Day 365. Note: based on clinical input, chest values of less than 30 mmHg and greater than 95 mmHg should not be used for the purpose of assigning chest value averages. Therefore, such values will not be considered for TcPO<sub>2</sub> ratio determination. Supplemental analyses using such values may be generated for exploratory purposes. The change in the TcPO<sub>2</sub> ratio from baseline will also be calculated. The TcPO<sub>2</sub> ratio and the change in TcPO<sub>2</sub> from baseline will be summarized by study visit and study arm using the method for continuous variables.

## 10.2.2.1 Imputation Methods of TCPO<sub>2</sub> Results for the ITT Population

For subjects without the efficacy endpoint (TCPO<sub>2</sub> change from baseline to any post baseline result), the following imputation methods will be applied:

- For missing Baseline TCPO<sub>2</sub>, assign the TCPO<sub>2</sub> score at Screening if the TCPO<sub>2</sub> score at Day 0 is missing.
- For any post baseline TCPO<sub>2</sub>, assign the post baseline TCPO<sub>2</sub> score prior to the missing post baseline TCPO<sub>2</sub> via the last observation carried forward (LOCF) method.

For subjects who had a major amputation or limb procedure carried out, the following imputation methods will be applied:

- For subjects with a major amputation, assign the TcPO<sub>2</sub> score prior to the amputation.
- For subjects with a limb salvage, assign the TcPO<sub>2</sub> score prior to the intervention.

## 10.2.3. HEMODYNAMIC ASSESSMENTS (ABI/TBI)

Hemodynamic assessments taken on the index limb and contra-lateral limb include the following:

- Resting Ankle Brachial-Index (ABI) measurements taken on both legs.
- Resting Toe Brachial-Index (TBI) measurements taken on toe of right and left foot.

Resting ABI and TBI and the change from baseline (= post-treatment – baseline) will be summarized by index/non-index limb, study visit, and treatment arm using the method for continuous variables. A value of 0 will be assigned if no pulse is reported. Same as the transcutaneous oxygen pressure measurements described in Section 10.2.2, the baseline value is the measurement taken at the Day-0 (Pre-Dose) Visit if the percent difference between the measurements taken at the Screening Visit and the Day-0 Visit is  $\leq 15\%$ . Otherwise, the baseline value is the average of the measurements taken at Screening and Day-0 Visits. The change in ABI and TBI from baseline will be summarized by study visit and study arm using the method for continuous variables. Supplemental analysis for exploratory purposes may be generated that does not consider subjects who have a baseline TBI/ABI between .9-1.3 mmHg.

## 10.2.3.1 Imputation Methods of ABI/TBI Results for the ITT Population

For subjects without the efficacy endpoint (ABI/TBI change from baseline to any post baseline result), the following imputation methods will be applied:

- For missing Baseline ABI/TBI, assign the ABI/TBI score at Screening if the ABI/TBI score score at Day 0 is missing.
- For any post baseline ABI/TBI, assign the post baseline ABI/TBI score prior to the missing post baseline ABI/TBI via the last observation carried forward (LOCF) method.

For subjects who had a major amputation or limb procedure carried out, the following imputation methods will be applied:

- For subjects with a major amputation, assign the ABI/TBI score prior to the amputation.
- For subjects with a limb salvage, assign the ABI/TBI score prior to the intervention.

#### 10.2.4. HIGH RESOLUTION MRA

The quantitative blood flow of the occluded target artery and the volumetric analysis of the newly developed artery will be recorded on a CRF for selected sites. The perfusion data at baseline, 6 months, and 9 months, and the change in perfusion from baseline to 6 and 9 months will be summarized descriptively using method for continuous variables at baseline, 6 months, and 9 months. The descriptive summaries will be provided by the independent laboratory. No statistical tests will be performed.

#### 10.2.5. Wound Healing and Ulcer Measurement

Based on photographs and measurements of ulcers, the length and width (in cm) of the ulcer will be recorded by the wound core lab. Additionally, the area of the open ulcer (in cm<sup>2</sup>) will be measured by the wound core lab. If an ulcer is determined to be 100% healed, the area of the ulcer will be set to 0. Descriptive statistics of the sum of ulcer areas and change from baseline will be performed by treatment arm and visit. The number of subjects with a 100% healed ulcer will be summarized by visit and treatment arm using the method for categorical variables.

## 10.2.6. QUALITY OF LIFE (VASCUQOL)

The VascuQoL contains five domains (activity, symptom, pain, emotion and social functioning). Each domain is scored on a scale from 1 to 7 based on the VascuQoL manual.

Scores will be assigned to responses according to the following table:

| VascuQoL<br>Question(s) | Score Assigned= Response |
|---|---|
| 1, 2, 5, 6, 7, 12, 13,<br>17, 19, 21, 23, 25 | 1= All of the time; 2= Most of the time; 3= Much of the time; 4= Some of the time; 5= A little of the time; 6= Hardly any of the time; 7= None of the time |
| 3, 8, 20 | 1= A very great deal of discomfort or distress; 2= A great deal of discomfort or distress; 3= A good deal of discomfort or distress; 4= A moderate amount of discomfort or distress; 5= Some discomfort or distress; 6= Very little discomfort or distress; 7= No discomfort or distress |
| 4 | 1= Total limited, couldn't exercise at all; 2= Extremely limited; 3= Very limited; 4= Moderately limited; 5= A little limited; 6= Only very slightly limited; 7= Not at all limited |
| 9 | 1= Not at all; 2= A little; 3= Somewhat; 4= Moderately; 5=A good deal; 6= A great deal; 7= A very great deal |
| 10 | 1= Total limited, couldn't walk at all; 2= Extremely limited; 3= Very limited; 4= Moderately limited; 5= A little limited; 6= Only very slightly limited; 7= Not at all limited |
| 11, 24 | 1= A very great deal; 2= A great deal; 3=A good deal; 4=<br>Moderately; 5= Somewhat; 6= A little; 7= Not at all |
| 14 | 1= Total limited, couldn't climb stairs at all; 2= Extremely limited; 3= Very limited; 4= Moderately limited; 5= A little limited; 6= Only very slightly limited; 7= Not at all limited |
| 15 | 1= Total limited, couldn't socialize at all; 2= Extremely limited; 3= Very limited; 4= Moderately limited; 5= A little limited; 6= Only very slightly limited; 7= Not at all limited |
| 16 | 1= Total limited, couldn't perform housework; 2= Extremely limited; 3= Very limited; 4= Moderately limited; 5= A little limited; 6= Only very slightly limited; 7= Not at all limited |
| 18 | 1= Severely limited; 2= Very limited; 3= Moderately limited; 4= Slightly limited; 5= Very slightly limited; 6= Hardly limited at all; 7=Not limited at all |
| 22 | 1= Total limited, couldn't go shopping at all 2= Extremely limited;<br>3= Very limited; 4= Moderately limited; 5= A little limited; 6=<br>Only very slightly limited; 7= Not at all limited |

The domain score is the total of the non-missing scores in the domain divided by the number of responded questions in the domain. The total King's College Hospital's VascuQol score is the total non-missing score divided by the total number of responded questions.

The following question numbers represent the various domains.

| Domain | VascuQoL Questions |
|-----------|------------------------------|
| Activity | 4, 9, 10, 14, 16, 18, 22, 24 |
| Symptom | 3, 5, 8, 17 |
| Pain | 1, 7, 13, 20 |
| Emotional | 2, 11, 12, 19, 21, 23, 25 |
| Social | 6, 15 |

Each QoL domain, the King's College Hospital's VascuQol score and each individual question will be summarized by treatment arm and study visit by the methods for continuous variables. Change from baseline will be also be summarized.

## 10.2.6.1 Imputation Methods of VASCUQOL Results for the ITT Population

For subjects without the efficacy endpoint (VASCUQOL change from baseline to any post baseline result), the following imputation methods will be applied:

- For missing Baseline VASCUQOL, assign the VASCUQOL score at Screening if the VASCUQOL score score at Day 0 is missing.
- For any post baseline VASCUQOL, assign the post baseline VASCUQOL score prior to the missing post baseline VASCUQOL via the last observation carried forward (LOCF) method.

For subjects who had a major amputation or limb procedure carried out, the following imputation methods will be applied:

- For subjects with a major amputation, assign the VASCUQOL score prior to the amputation.
- For subjects with a limb salvage, assign the VASCUQOL score prior to the intervention.

## 10.2.7. Amputation and Mortality Rate

The rates of amputation, limb salvage and mortality will be analyzed for all treated subjects per actual treatment using the method for time-to-event variables. The probability of being event-free at 6 and 12 months will be summarized for each treatment arm and compared *vs.* Placebo using a Log Rank test.

The duration of time to amputation will be defined as the number of days between the day of amputation – the first dose date + 1. If a subject does not report amputation, then the date that the subject will be censored at the date of study discontinuation. If the date of study of discontinuation is not available, then the subject's censor date will be the last known visit the subject attended. The same calculation will be repeated for limb salvage and mortality (time to death).

## 10.2.8. Rutherford Classification

The Rutherford Classification measurement (which characterizes peripheral arterial disease severity using a discrete 7 point scale from 0-6) and change from baseline will be summarized at each visit by treatment arm using method for continuous variables.

## 10.2.8.1 Imputation Methods of Rutherford Results for the ITT Population

For subjects without the efficacy endpoint (Rutherford Classification change from baseline to any post baseline result), the following imputation methods will be applied:

- For missing Baseline Rutherford Classification, assign the Rutherford Classification score at Screening if the Rutherford Classification score score at Day 0 is missing.
- For any post baseline Rutherford Classification, assign the post baseline Rutherford Classification score prior to the missing post baseline Rutherford Classification via the last observation carried forward (LOCF) method.

For subjects who had a major amputation or limb procedure carried out, the following imputation methods will be applied:

• For subjects with a major amputation, assign the Rutherford Classification score prior to the amputation.

• For subjects with a limb salvage, assign the Rutherford Classification score prior to the intervention.

#### 10.3. Baseline Values

Unless specified otherwise, the baseline value for each variable is the last non-missing value recorded at the last visit on or before start of dosing. In most cases, baseline values are expected to be based on the assessment collected at the Day 0 (Pre-Dose) visit.

## 10.4. Multiplicity Adjustments

Pairwise comparisons using Dunnett's test adjust for multiple comparisons. Otherwise, there will be no adjustments for multiple comparisons or interim analyses.

#### 11. SAFETY ANALYSES

All subjects who received study drug will be included in the safety analyses, analyzed according to the study treatment actually received.

## 11.1. Study Drug Exposure

Study drug exposure will be summarized descriptively by treatment arm for Day 0, Day 14, Day 28 and Day 42. Categorical variables to be summarized using counts and percentages include "Was dose administered?" (Yes, No), the zone of the dose administration (I, II, III, IV) and "Was the total volume (8 mL) administered?" (Yes, No). In addition, the elapsed time of study drug administered (continuous variable) will be summarized in minutes using descriptive statistics.

#### 11.2. Adverse Events

All adverse event summaries will be restricted to Treatment Emergent Adverse Events (TEAE), which are defined as those AEs that occurred on or after first dosing date and those existing AEs that worsened during the study. Verbatim terms on case report forms

will be mapped to preferred terms and system organ classes using the MedDRA dictionary (version 14.0).

Each adverse event summary will be displayed by treatment arm. Summaries that are displayed by system organ class and preferred terms will be ordered by descending order of incidence of system organ class and preferred term within each system organ class. The number of subjects experiencing a particular event, the percentage of subjects experiencing the event will be presented. The total number of events will be presented for a select set of summaries. The following summaries will be created:

- TEAE by MedDRA system organ class and preferred term;
- TEAE by MedDRA system organ class, preferred term, and maximum severity. At each level of subject summarization a subject is classified according to the highest severity if the subject reported one or more events. AEs with missing severity will be considered severe for this summary;
- TEAE by MedDRA system organ class, preferred term, and closest relationship to study drug (Related/Unrelated). At each level of subject summarization a subject is classified according to the closest relationship if the subject reported one or more events. AEs with a missing relationship will be considered related for this summary; Events classified as 'possibly', 'probably' or 'definitely' will be considered 'related';
- Serious TEAEs by MedDRA system organ class and preferred term.

## 11.3. Clinical Laboratory Evaluation

Shift tables (i.e., low-normal-high at baseline versus low-normal-high at follow-up in a 3-by-3 contingency table) will be provided to assess changes in laboratory values from baseline to each planned post-baseline visit. The counts and percentage of subjects with each of the 9 possible "shift" outcomes will be calculated by treatment arm.

## 11.4. Vital Signs

Vital signs and change from baseline will be summarized descriptively at each visit by treatment arm. Changes from baseline will also be summarized. Baseline is defined as the last non-missing value prior to first dose of study drug.

## 11.5. Retinal Fundoscopy

A retinal fundoscopy of each eye will be performed at Screening and at 12 Months. In the case of an early withdrawal, a retinal fundoscopy may be performed prior to 12 Months. Each eye will be given one of the following assignments: Normal, Abnormal-Not Clinically Significant, and Abnormal-Clinically Significant. Shift tables will be provided to assess changes in retinal fundoscopy. Shift tables will summarize changes from Screening to 12 Months. If a 12 Month assessment was not performed, the last post-baseline assessment reported will be used. For each of the three treatment groups, counts and percentage of subjects will be calculated for each of the 9 possible "shift" outcomes.

## 11.6. Injection Site Reaction

Assessments of the existence of an injection site reaction (Yes or No) are planned for Day 0 (post-dose), Day 14 (pre and post dose), Day 28 (pre and post dose), Day 42 (pre and post dose) and Day 49. The number and percentage of subjects with and without an injection site reaction will be summarized descriptively by treatment arm and study visit.

#### 11.7. Prior and Concomitant Medications

Verbatim terms on case report forms will be mapped to Anatomical/Therapeutic/Chemical (ATC) Level 4 categories and Drug Reference Names using the World Health Organization (WHO) dictionary (March 1, 2011).

Prior medications are those medications taken within 30 days prior to the initial dose of study drug. Concomitant medications are those medications taken after the initial dose of study drug. Prior and concomitant medications will be summarized for each treatment by WHO ATC class and medication name. These summaries will present the number and percentage of subjects using each medication. Subjects may have more than one medication per ATC category and medication. At each level of subject summarization, a subject is counted once if he/she reported one or more medications at that level. Each summary will be ordered by descending order of incidence of ATC class and medication within each ATC class.

## 11.8. Interim Analyses

An interim analysis of key safety data will be performed when approximately half of the subjects (n=25) have 6 month data. The primary objective of this analysis will be to evaluate the accumulating data for an unacceptably high frequency of negative clinical outcomes in either active treatment arm. An independent data safety monitoring board (DSMB) will review a limited set of un-blinded tables and listings, including all reported SAEs. There will be no adjustment for multiple testing because the results of the interim analysis will not be used to declare the study a success.

## APPENDIX A: LIST OF TABLES AND LISTINGS

# **List of Tables**

| Table | |
|---|---|
| Number | Table Description |
| 1 | Subject Disposition |
| 2.1 | Demographic and Baseline Characteristics (ITT Populations) |
| 2.2 | Demographic and Baseline Characteristics (Safety Populations) |
| 2.3 | Demographic and Baseline Characteristics (Per-Protocol Populations) |
| 3 | Medical History (Safety Population) |
| 4 | Peripheral Vascular Disease Intervention History (Safety Population) |
| 5.1.1 | Visual Analogue Scale for Pain (Per-Protocol Population) |
| 5.1.2 | Visual Analogue Scale for Pain (ITT Population) |
| 5.2.1 | Visual Analogue Scale for Pain- Percent (%) Change from Baseline |
| | (Per-Protocol Population) |
| 5.2.2 | Visual Analogue Scale for Pain- Percent (%) Change from Baseline (ITT |
| | Population) |
| 5.3.1.1 | Visual Analogue Scale for Pain at 9 Months by Sex (Per-Protocol |
| | Population) |
| 5.3.1.2 | Visual Analogue Scale for Pain at 9 Months by Sex (ITT Population) |
| 5.3.2.1 | Visual Analogue Scale for Pain at 9 Months by Renal Dysfunction |
| | (Per-Protocol Population) |
| 5.3.2.2 | Visual Analogue Scale for Pain at 9 Months by Renal Dysfunction (ITT |
| | Population) |
| 5.3.3.1 | Visual Analogue Scale for Pain at 9 Months by Diabetes (Per-Protocol |
| | Population) |
| 5.3.3.2 | Visual Analogue Scale for Pain at 9 Months by Diabetes (ITT Population) |
| 5.4.1 | Categorical Analysis of Visual Analogue Scale for Pain (Per-Protocol |
| 5.4.2 | Population) |
| 5.4.2 | Categorical Analysis of Visual Analogue Scale for Pain (ITT Population) |
| 6.1.1.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Anterior Calf |
| (112 | (Per-Protocol Population) |
| 6.1.1.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Anterior Calf (ITT |
| | Population) |

| (121 | Tanasata and Carres Burney Annual Tanasa Tanasa Bartai a Calif |
|---|---|
| 6.1.2.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Posterior Calf (Per-Protocol Population) |
| 6.1.2.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Posterior Calf (ITT |
| 0.1.2.2 | Population) |
| 6121 | i |
| 6.1.3.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Dorsum Foot |
| 6122 | (Per-Protocol Population) |
| 6.1.3.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Dorsum Foot (ITT |
| | Population) |
| 6.1.4.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Chest |
| | (Per-Protocol Population) |
| 6.1.4.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> - Chest (ITT |
| | Population) |
| 6.2.1.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> Ratio - Anterior Calf |
| | (Per-Protocol Population) |
| 6.2.1.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> Ratio - Anterior Calf |
| | (ITT Population) |
| 6.2.2.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> Ratio - Posterior |
| | Calf (Per-Protocol Population) |
| 6.2.2.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> Ratio - Posterior |
| | Calf (ITT Population) |
| 6.2.3.1 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> Ratio- Dorsum Foot |
| | (Per-Protocol Population) |
| 6.2.3.2 | Transcutaneous Oxygen Pressure Assessment- TcPO <sub>2</sub> Ratio - Dorsum Foot |
| | (ITT Population) |
| 7.1.1 | Ankle Brachial-Index – Index Leg (Per-Protocol Population) |
| 7.1.2 | Ankle Brachial-Index – Index Leg (ITT Population) |
| 7.2.1 | Ankle Brachial-Index – Non-Index Leg (Per-Protocol Population) |
| 7.2.2 | Ankle Brachial-Index – Non-Index Leg (ITT Population) |
| 8.1.1 | Toe Brachial-Index – Index Leg (Per-Protocol Population) |
| 8.1.2 | Toe Brachial-Index – Index Leg (ITT Population) |
| 8.2.1 | Toe Brachial-Index – Non-Index Leg (Per-Protocol Population) |
| 8.2.2 | Toe Brachial-Index – Non-Index Leg (ITT Population) |
| 9.1.1 | Wound Area (Per-Protocol Population) |
| 9.1.2 | Wound Area (ITT Population) |
| 9.2.1 | Categorical Analysis of Wound Healing (Per-Protocol Population) |
| 9.2.2 | Categorical Analysis of Wound Healing (ITT Population) |
| 10.1.1 | VascuQoL – Activity (Per-Protocol Population) |

| 10.1.2 | VascuQoL – Activity (ITT Population) |
|---|---|
| 10.1.2 | VascuQoL – Activity (11 1 Topulation) VascuQoL – Symptom (Per-Protocol Population) |
| 10.2.1 | VascuQoL – Symptom (Fet-Flotocol Fopulation) VascuQoL – Symptom (ITT Population) |
| 10.2.2 | VascuQoL – Symptom (111 Fopulation) VascuQoL – Pain (Per-Protocol Population) |
| | · |
| 10.3.2 | VascuQoL – Pain (ITT Population) |
| 10.4.1 | VascuQoL – Emotional (Per-Protocol Population) |
| 10.4.2 | VascuQoL – Emotional (ITT Population |
| 10.5.1 | VascuQoL – Social (Per-Protocol Population) |
| 10.5.2 | VascuQoL – Social (ITT Population) |
| 10.6.1 | VascuQoL – Total (Per-Protocol Population) |
| 10.6.2 | VascuQoL – Total (ITT Population) |
| 10.7.1 | VascuQoL- By Individual Question (Per-Protocol Population) |
| 10.7.2 | VascuQoL- By Individual Question (ITT Population) |
| 11.1.1 | Amputation – Event-Free Probability (Per-Protocol Population) |
| 11.1.2 | Amputation – Event-Free Probability (ITT Population) |
| 11.2.1 | Limb Salvage – Event-Free Probability (Per-Protocol Population) |
| 11.2.2 | Limb Salvage – Event-Free Probability (ITT Population) |
| 11.3.1 | Mortality – Event-Free Probability (Per-Protocol Population) |
| 11.3.2 | Mortality – Event-Free Probability (ITT Population) |
| 12.1 | Rutherford Classification of Disease Severity (Per-Protocol Population) |
| 12.2 | Rutherford Classification of Disease Severity (ITT Population) |
| 13 | Study Drug Exposure(Safety Population) |
| 14 | Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| 15 | Treatment Emergent Adverse Events by Maximum Severity (Safety |
| | Population) |
| 16 | Treatment Emergent Adverse Events by Relationship to Study Drug |
| | (Safety Population) |
| 17 | Treatment Emergent Serious Adverse Events by System Organ Class and |
| | Preferred Term (Safety Population) |
| 18 | Hematology –Shift from Baseline (Safety Population) |
| 19 | Serum Chemistry –Shift from Baseline (Safety Population) |
| 20 | Vital Signs – Parameter # (Safety Population) |
| 21 | Retinal Fundoscopy- Shift from Baseline (Safety Population) |
| 22 | Injection Site Reaction (Safety Population) |
| 23 | Prior and Concomitant Medications (Safety Population) |
| | (=) |

# **List of Figures**

| Figure | |
|--------|--------------------------------------|
| Number | Figure Description |
| 1 | Amputation- Event Free Probability |
| 2 | Limb Salvage- Event Free Probability |
| 3 | Mortality- Event Free Probability |

# **List of Listings**

| Listing | |
|---------|-------------------------------------------------------------|
| Number | Listing Description |
| 1 | Subject Disposition |
| 2 | Protocol Deviation |
| 3 | Eligibility Criteria |
| 4 | Demographics and Baseline Characteristics |
| 5 | Medical History |
| 6 | Peripheral Vascular Disease Intervention History |
| 7 | Physical Examination at Screening |
| 8 | Chest X-Ray/ CT Scan |
| 9 | Infection Screening |
| 10 | Urine Pregnancy Test |
| 11 | Mammogram |
| 12 | PAP Smear |
| 13 | 12-Lead Electrocardiogram |
| 14 | Fecal Occult Blood Test |
| 15 | Gastroscopy |
| 16 | Colonoscopy |
| 17 | Tumor Markers |
| 18 | Visual Analog Scale (VAS) for Pain |
| 19 | Resting Transcutaneous Oxygen Pressure (TcPO2) Measurements |
| 20 | Resting Ankle Brachial Index (ABI) Measurements |
| 21 | Resting Toe Brachial Index (TBI) Measurements |
| 22 | Ulcer and Wound Assessment/ Skin Condition Assessment |
| 23 | Ulcer Assessment |
| 24 | Vascular Quality of Life (VascuQoL) |
| 25 | High Resolution Magnetic Resonance Angiography (MRA) |
| 26 | Rutherford Classification |
| 27 | Study Drug Administration |
| 28 | Adverse Events |
| 29 | Serious Adverse Events |
| 30 | Hematology |
| 31 | Serum Chemistry |

| 32 | Urinalysis |
|----|--------------------------------------|
| 33 | Vital Signs |
| 34 | Copies of VM202 in Whole Blood |
| 35 | Serum Hepatocyte Growth Factor (HGF) |
| 36 | Eye Examination- Retinal Fundoscopy |
| 37 | Injection Site Reaction |
| 38 | Prior and Concomitant Medications |
| 39 | Prior and Concomitant Procedures |
| 40 | Death Report |

# **APPENDIX B: TABLE LAYOUTS**

**Protocol Number: VMCLI-II-09-002** 

#### Table 1 **Subject Disposition** All Subjects

| | Placebo | VM202- 8 mg | VM202- 16 mg |
|---|---|---|---|
| Subjects Enrolled | n (Overall) | | |
| ITT Population [1] | n | n | n |
| Safety Population [2] | n (%) | n (%) | n (%) |
| Per-Protocol Population [3] | n (%) | n (%) | n (%) |
| Received All Planned Doses of VM202? | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Last Visit Attended | | | |
| Any Visit Prior to Visit- Day 0 | n (%) | n (%) | n (%) |
| Visit- Day 0 | n (%) | n (%) | n (%) |
| Visit- Day 14 | n (%) | n (%) | n (%) |
| Visit- Day 28 | n (%) | n (%) | n (%) |
| Visit- Day 42 | n (%) | n (%) | n (%) |
| Visit- Day 49 | n (%) | n (%) | n (%) |
| Visit- Day 90 | n (%) | n (%) | n (%) |
| Visit- 6 Months | n (%) | n (%) | n (%) |
| Visit- 9 Months | n (%) | n (%) | n (%) |
| Visit- 12 Months | n (%) | n (%) | n (%) |
| Completed Study? | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |

Page 1 of 2

Note: Percentages based on number of subjects in the ITT population.

[1] All subjects who were randomized regardless of whether treatment was received.

[2] All subjects who received at least one dose of study drug.

[3] All subjects who received the correct dose of study drug medication, have the 9-month VAS assessment, and do not have any protocol violations or major deviations. path\t\_program.sas date

**Protocol Number: VMCLI-II-09-002** 

Table 1 **Subject Disposition** All Subjects

| | Placebo | VM202- 8 mg | VM202- 16 mg |
|---|---|---|---|
| Primary Reason for Discontinuation | | | |
| Screen failure | n (%) | n (%) | n (%) |
| Lost to Follow-up | n (%) | n (%) | n (%) |
| Adverse Event | n (%) | n (%) | n (%) |
| Non-compliance | n (%) | n (%) | n (%) |
| Subject withdrew consent | n (%) | n (%) | n (%) |
| Principal Investigator decision | n (%) | n (%) | n (%) |
| Subject requires intervention for treatment of acute limb ischemia | n (%) | n (%) | n (%) |
| Death | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |

Page 2 of 2

Note: Percentages based on number of subjects in the ITT population.

[1] All subjects who were randomized regardless of whether treatment was received.

[2] All subjects who received at least one dose of study drug.

[3] All subjects who received the correct dose of study drug medication, have the 9-month VAS assessment, and do not have any protocol violations or major deviations. path\t program.sas date

ViroMed Co., Ltd. **Protocol Number: VMCLI-II-09-002** 

Table 2.1 **Demographic and Baseline Characteristics ITT Population** 

| | Placebo (N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) | <i>p</i> -value |
|---|---|---|---|---|
| | (IN- ) | (IN- ) | (N- ) | p-value |
| Age (years) [1] | | | | |
| N | n | n | n | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | x.xxxx [2] |
| Median | xx.x | xx.x | xx.x | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Sex | | | | x.xxxx <sup>[3]</sup> |
| Male | n (%) | n (%) | n (%) | |
| Female | n (%) | n (%) | n (%) | |
| Race | | | | x.xxxx <sup>[3]</sup> |
| Caucasian | n (%) | n (%) | n (%) | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) | |
| Black or African American | n (%) | n (%) | n (%) | |
| Asian | n (%) | n (%) | n (%) | |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) | |
| Hispanic or Latino | n (%) | n (%) | n (%) | |
| Other | n (%) | n (%) | n (%) | |
| Height (in) | | | | |
| N | n | n | n | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | x.xxxx [2] |
| Median | xx.x | xx.x | xx.x | |
| Min, Max | XX, XX | XX, XX | XX, XX | |

<sup>[1]</sup> Age calculated by determining the number of years between the date of informed consent and the date of birth. [2] *P*-value tests for treatment difference using a one-way analysis of variance (ANOVA).

path\t\_program.sas date

Programmer note Table 2.2 will be identical to Table 2.1 for the Safety Population. Table 2.3 will be identical to Table 2.1 for the Per-Protocol Population.

<sup>[3]</sup> P-value tests for treatment difference using a Fisher's exact test.
Table 2.1 **Demographic and Baseline Characteristics ITT Population** 

| | Placebo (N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) | <i>p</i> -value |
|---|---|---|---|---|
| | (11) | (11) | (11) | p value |
| Weight (lb) | | | | |
| N | n | n | n | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | x.xxxx [2] |
| Median | XX.X | xx.x | xx.x | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Does the subject have diabetes mellitus? | | | | x.xxxx [3] |
| Yes | n (%) | n (%) | n (%) | |
| No | n (%) | n (%) | n (%) | |
| Does the subject have renal dysfunction? | | | | x.xxxx [3] |
| Yes | n (%) | n (%) | n (%) | |
| No | n (%) | n (%) | n (%) | |

<sup>[1]</sup> Age calculated by determining the number of years between the date of informed consent and the date of birth.
[2] P-value tests for treatment difference using a one-way analysis of variance (ANOVA).
[3] P-value tests for treatment difference using a Fisher's exact test.

path\t\_program.sas date time

Programmer note Table 2.2 will be identical to Table 2.1 for the Safety Population. Table 2.3 will be identical to Table 2.1 for the Per-Protocol Population.

Protocol Number: VMCLI-II-09-002

Table 3 Medical History Safety Population

| | Placebo | VM202- 8 mg | VM202- 16 mg |
|----------------------------|---------|-------------|--------------|
| Body System | (N= ) | (N= ) | (N= ) |
| Respiratory | n (%) | n (%) | n (%) |
| Cardiovascular | n (%) | n (%) | n (%) |
| Gastrointestinal | n (%) | n (%) | n (%) |
| Hepatic | n (%) | n (%) | n (%) |
| Endocrine/Metabolic | n (%) | n (%) | n (%) |
| Central Nervous System | n (%) | n (%) | n (%) |
| Hematopoietic/Lymphatic | n (%) | n (%) | n (%) |
| Dermatological | n (%) | n (%) | n (%) |
| Musculoskeletal | n (%) | n (%) | n (%) |
| Genitourinary/Reproductive | n (%) | n (%) | n (%) |
| Psychiatric | n (%) | n (%) | n (%) |
| Alcohol/Drug Abuse | n (%) | n (%) | n (%) |
| Drug Allergy | n (%) | n (%) | n (%) |
| Non-Drug Allergy | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Protocol Number: VMCLI-II-09-002

Table 4
Peripheral Vascular Disease Intervention History
Safety Population

| | Placebo | VM202- 8 mg | VM202- 16 mg |
|---------------------------|---------|-------------|--------------|
| Intervention | (N= ) | (N= ) | (N= ) |
| PTA | n (9/) | - (0/) | m (0/) |
| | n (%) | n (%) | n (%) |
| Peripheral bypass | n (%) | n (%) | n (%) |
| Amputation above the knee | n (%) | n (%) | n (%) |
| Amputation below the knee | n (%) | n (%) | n (%) |
| Atherectomy | n (%) | n (%) | n (%) |
| Surgical bypass | n (%) | n (%) | n (%) |
| Endarterectomy | n (%) | n (%) | n (%) |
| Thrombectomy | n (%) | n (%) | n (%) |
| Stent placement | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |

path\t\_program.sas date time


**Protocol Number: VMCLI-II-09-002** 

**Table 5.1.1** Visual Analogue Scale for Pain (mm) **Per-Protocol Population** 

| | Placebo | | | | VM202- 10 | |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | |
| N N | | | | | | |
| Mean (SD) | n<br> | | n | | n<br>···································· | |
| Median | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | |
| Day 14 | | | | | | |
| Ň | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | () | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| 7370 Of for Est Michiel Silicitation | | | | (AA.A, A.AA) | | (AA.A, A.AA) |
| Overall p-value for Treatment Differences | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Dunnett's test) | | | | X.XXXX | | X.XXXX |
| Baseline vs. Day 14 (Paired t-test) | | X.XXXX | | X.XXXX | | X.XXXX |
| Model 2 [4] | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | x.xxxx |
| Pairwise <i>p</i> -value vs. Placebo (Wilcoxon Rank Sum test) | | | | x.xxxx | | X.XXXX<br>X.XXXX |
| Baseline vs. Day 14 (Wilcoxon Signed Rank test) | | x.xxxx | | X.XXXX | | X.XXXX |
| Dascille vs. Day 14 (Wilcoxoll Signed Rallk test) | | Λ.ΑΧΧΧ | | Λ.ΛΧΧΧ | | Λ.ΑΧΧΧ |

<sup>[1]</sup> Baseline defined as the last non-missing value prior to first dose of study drug.
[2] Change = Change from Baseline

Programmer Note Repeat for all available time points, Day 14, Day 28, Day 42, Day 90, 6mo, 9mo, and 12mo.

Programmer Note Tables 5.1.2 will be identical to Table 5.1.1 for the ITT Population using imputation rules specified in Section 10.1.2 of the Statistical Analysis Plan.

Change – Change from Baseline

[3] One –way analysis of variance (ANOVA) with treatment groups as a factor.

[4] Nonparametric tests for differences across a one-way classification of treatment. path\t\_program.sas date

**Protocol Number: VMCLI-II-09-002** 

**Table 5.2.1** Visual Analogue Scale for Pain- Percent (%) Change from Baseline **Per-Protocol Population** 

| | Placebo | VM202- 8 mg | VM202-16 mg |
|---|---|---|---|
| | (N= ) | (N= ) | (N= ) |
| | Change <sup>[2]</sup> | Change [2] | Change <sup>[2]</sup> |
| Devil A Deview (0/) Character Paralline [1] | | | |
| Day 14- Percent (%) Change from Baseline [1] | | | |
| N<br>W (GP) | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx |
| Comparison vs. Placebo | | | |
| Model 1 [3] | | | |
| LS Means (SE) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| LS Mean Differences (SE) | ` ′ | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI for LS Mean Differences | | (xx.x, x.xx) | (xx.x, x.xx) |
| Overall p-value for Treatment Differences | | | x.xxxx |
| Pairwise p-value vs. Placebo (Dunnett's test) | | x.xxxx | x.xxxx |
| Baseline vs. Day 14 (Paired t-test) | x.xxxx | X.XXXX | x.xxxx |
| Model 2 [4] | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | x.xxxx |
| Pairwise p-value vs. Placebo (Wilcoxon Rank Sum test) | | x.xxxx | X.XXXX |
| 1 | V VVVV | | |
| Baseline vs. Day14 (Wilcoxon Signed Rank test) | X.XXXX | X.XXXX | X.XXXX |

Programmer Note Repeat for all available time points, Day14, Day 28, Day 42, Day 90, 6mo, 9mo, and 12mo.

Programmer Note Tables 5.2.2 will be identical to Table 5.2.1 for the ITT Population using imputation rules specified in Section 10.1.2 of the Statistical Analysis Plan.

Baseline defined as the last non-missing value prior to first dose of study drug.
 Change = Change from Baseline
 One -way analysis of variance (ANOVA) with treatment groups as a factor.
 Nonparametric test for differences across a one-way classification of treatment. path\t program.sas date time

ViroMed Co., Ltd. Page 1 of 1

Protocol Number: VMCLI-II-09-002

### **Table 5.3.1.1** Visual Analogue Scale for Pain (mm) at 9 Months by Sex **Per-Protocol Population**

| | Placebo (N= ) | | | | VM202- 1 | |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| All Subjects: Model 1 [3] Overall <i>p</i> -value for Treatment-by-Sex Factor | | | | | | x.xxxx |
| Model 2 <sup>[4]</sup> LS Means (SE) LS Mean Differences (SE) 95% CI for LS Mean Differences Pairwise <i>p</i> -value <i>vs.</i> Placebo (Dunnett's t-test) | | xx.x (xx.x) | | xx.x (xx.x)<br>xx.x (xx)<br>(xx.x, x.xx)<br>x.xxxx | | xx.x (xx.x)<br>xx.x (xx)<br>(xx.x, x.xx)<br>x.xxxx |

<sup>[1]</sup> Baseline defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programmer Note Tables 5.3.1.2 will be identical to Table 5.3.1.1 for the ITT Population using imputation rules specified in Section 10.1.2 of the Statistical Analysis Plan. Programmer Note Table 5.3.2 and Table 5.3.3 will be identical to Table 5.3.1, except Renal Dysfunction and Diabetes will be used as factors instead of sex, respectively.

<sup>[2]</sup> Change = Change from Baseline

<sup>[3]</sup> Analysis of variance (ANOVA) with treatment group, sex and treatment-by-sex interaction as factors.
[4] Analysis of variance (ANOVA) with treatment group and sex as factors.
[5] One –way analysis of variance (ANOVA) with treatment groups as a factor.

<sup>[6]</sup> Nonparametric test for differences across a one-way classification of treatment.


**Protocol Number: VMCLI-II-09-002** 

ViroMed Co., Ltd.

**Table 5.3.1.1** Visual Analogue Scale for Pain (mm) at 9 Months by Sex **Per-Protocol Population** 

| | Placebo (N= ) | | VM202- 8 mg (N= ) | | VM202- 16 mg (N= ) | |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| V.1 | | | | | | |
| Males: Baseline [1] | | | | | | |
| N | _ | | | | _ | |
| Mean (SD) | n<br>xx.x (xx.xx) | | n<br>vv v (vv vv) | | n<br>vv v (vv vv) | |
| Median | ` / | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | |
| 9 Months | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Model 3 [5] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | , , | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| Overall <i>p</i> -value for Treatment Differences | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Dunnett's test) | | | | x.xxxx | | X.XXXX |
| Baseline vs. 9 Months (Paired t-test) | | x.xxxx | | X.XXXX | | X.XXXX |
| Baseline vs. 7 Wollans (1 and t-test) | | Λ.ΛΛΛΛ | | Α.ΑΑΑΑ | | Λ.ΛΛΛΛ |
| Model 4 [6] | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Wilcoxon Rank Sum test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 9 Months (Wilcoxon Signed Rank test) | | x.xxxx | | x.xxxx | | x.xxxx |

<sup>[1]</sup> Baseline defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date

Programmer Note Tables 5.3.1.2 will be identical to Table 5.3.1.1 for the ITT Population using imputation rules specified in Section 10.1.2 of the Statistical Analysis Plan. Programmer Note Table 5.3.2 and Table 5.3.3 will be identical to Table 5.3.1, except Renal Dysfunction and Diabetes will be used as factors instead of sex, respectively

<sup>[2]</sup> Change = Change from Baseline

Analysis of variance (ANOVA) with treatment group, sex and treatment-by-sex interaction as factors.

Analysis of variance (ANOVA) with treatment group and sex as factors.

Done—way analysis of variance (ANOVA) with treatment groups as a factor.

Nonparametric test for differences across a one-way classification of treatment. time

**Protocol Number: VMCLI-II-09-002** 

ViroMed Co., Ltd.

**Table 5.3.1.1** Visual Analogue Scale for Pain (mm) at 9 Months by Sex **Per-Protocol Population** 

| | Placebo (N= ) | | VM202- 8 mg (N= ) | | VM202- 10 | 6 mg (N= ) |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Females: | | | | | | |
| Baseline [1] | | | | | | |
| N | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| 9 Months | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx |
| Model 3 <sup>[5]</sup> | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | ` ′ | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| Overall <i>p</i> -value for Treatment Differences | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Dunnett's test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 9 Months (Paired t-test) | | X.XXXX | | X.XXXX | | x.xxxx |
| Model 4 <sup>[6]</sup> | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Wilcoxon Rank Sum test) | | | | x.xxxx | | X.XXXX |
| Baseline vs. 9 Months (Wilcoxon Signed Rank test) | | x.xxxx | | x.xxxx | | x.xxxx |

<sup>[1]</sup> Baseline defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programmer Note Tables 5.3.1.2 will be identical to Table 5.3.1.1 for the ITT Population using imputation rules specified in Section 10.1.2 of the Statistical Analysis Plan. Programmer Note Table 5.3.2 and Table 5.3.3 will be identical to Table 5.3.1, except Renal Dysfunction and Diabetes will be used as factors instead of sex, respectively

<sup>[2]</sup> Change = Change from Baseline

Change – Change from Baseline

[3] Analysis of variance (ANOVA) with treatment group, sex and treatment-by-sex interaction as factors.

[4] Analysis of variance (ANOVA) with treatment group and sex as factors.

[5] One –way analysis of variance (ANOVA) with treatment groups as a factor.

[6] Nonparametric test for differences across a one-way classification of treatment.

**Protocol Number: VMCLI-II-09-002** 

**Table 5.4.1** Categorical Analysis of Visual Analogue Scale for Pain (mm) **Per-Protocol Population** 

| | Placebo (N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| Baseline [1] | | | |
| 0-4 mm | n (%) | n (%) | n (%) |
| 5-44 mm | n (%) | n (%) | n (%) |
| 45-74 mm | n (%) | n (%) | n (%) |
| 75-100 mm | n (%) | n (%) | n (%) |
| Pairwise <i>p</i> -value vs. Placebo [2] | . , | .xxxx | .xxxx |
| Day 14 | | | |
| 0-4 mm | n (%) | n (%) | n (%) |
| 5-44 mm | n (%) | n (%) | n (%) |
| 45-74 mm | n (%) | n (%) | n (%) |
| 75-100 mm | n (%) | n (%) | n (%) |
| Pairwise <i>p</i> -value <i>vs</i> . Placebo <sup>[2]</sup> | | .xxxx | .xxxx |

path\t\_program.sas date

Programmer Note Repeat for all available time points, Day14, Day 28, Day 42, Day 90, 6mo, 9mo, and 12mo.

Programmer Note Tables 5.4.2 will be identical to Table 5.4.1 for the ITT Population using imputation rules specified in Section 10.1.2 of the Statistical Analysis Plan.

Note: Only subjects with ulcers at baseline are considered for analysis.  $^{[1]}$  Baseline defined as the last non-missing value prior to first dose of study drug.  $^{[2]}$  Pairwise p-value tests for treatment group difference using CMH test (Row Mean Scores).

**Table 6.1.1.1** Transcutaneous Oxygen Pressure Assessment- TcPO2 (mmHg) - Anterior Calf **Per-Protocol Population** 

| | Placebo<br>Result | (N= )<br>Change [2] | VM202- 8<br>Result | mg (N= )<br>Change <sup>[2]</sup> | VM202- 1<br>Result | 6 mg (N= )<br>Change <sup>[2]</sup> |
|---|---|---|---|---|---|---|
| Baseline [1] | | | | | | |
| N | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | |
| 6 Months | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | ` / | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| Overall <i>p</i> -value for Treatment Differences | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Dunnett's test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 6 Months (Paired t-test) | | x.xxxx | | x.xxxx | | x.xxxx |
| Model 2 [4] | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Wilcoxon Rank Sum test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 6 Months (Wilcoxon Signed Rank test) | | X.XXXX | | x.xxxx | | x.xxxx |

Baseline value is the ratio taken at the Day 0 (Pre-Dose) Visit if the percent difference (=|Day 0 - Screening $\times$ 100%) between the ratios taken at the Screening Visit and the Day-0 Visit is  $\leq$  15%. Otherwise, the baseline value is the average of the ratios at Screening and Day 0 Visits.

Programmer Note Repeat for all available time points, 6mo, 9mo and 12mo.

Programmer Note Tables 6.1.1.2 will be identical to Table 6.1.1.1 for the ITT Population using imputation rules specified in Section 10.2.2 of the Statistical Analysis Plan.

Programmer Note Tables 6.1.2, 6.1.3 and 6.1.4 will be identical to Table 6.1.1 for the Posterior Calf, Dorsum Foot and Chest.

<sup>[2]</sup> Change = Change from Baseline

One –way analysis of variance (ANOVA) with treatment groups as a factor.

<sup>[4]</sup> Nonparametric tests for differences across a one-way classification of treatment. path\t program.sas date time

Page x of x

Protocol Number: VMCLI-II-09-002

ViroMed Co., Ltd.

**Table 6.2.1.1** Transcutaneous Oxygen Pressure Assessment-TcPO2 Ratio - Anterior Calf **Per-Protocol Population** 

| | Placebo | Placebo (N= ) | | VM202- 8 mg (N= ) | | 6 mg (N= ) |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | |
| N N | | | | | | |
| Mean (SD) | n<br>vv v (vv vv) | | n<br>vv v (vv vv) | | n<br>vv v (vv vv) | |
| Median | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | |
| 6 Months | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| ye we critical and management | | | | (,) | | (111111, 111111) |
| Overall p-value for Treatment Differences | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Dunnett's test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 6 Months (Paired t-test) | | x.xxxx | | x.xxxx | | x.xxxx |
| Model 2 [4] | | | | | | |
| Overall p-value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | X.XXXX |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Wilcoxon Rank Sum test) | | | | X.XXXX | | X.XXXX |
| Baseline vs. 6 Months (Wilcoxon Signed Rank test) | | x.xxxx | | X.XXXX | | x.xxxx |

Note: TcPO<sub>2</sub> Ratio = Anterior Calf TcPO<sub>2</sub> / Chest TcPO<sub>2</sub>.

Programmer Note Repeat for all available time points, 6mo, 9mo and 12mo.

Programmer Note Tables 6.2.1.2 will be identical to Table 6.2.1.1 for the ITT Population using imputation rules specified in Section 10.2.2 of the Statistical Analysis Plan.

Programmer Note Tables 6.2.2 and 6.2.3 will be identical to Table 6.2.1 for the TcPO2 Ratios- Posterior Calf and Dorsum Foot.

Baseline value is the ratio taken at the Day 0 (Pre-Dose) Visit if the percent difference (=|Day 0 - Screening/Screening×100%) between the ratios taken at the Screening Visit and the Day-0 Visit is  $\leq$ 15%. Otherwise, the baseline value is the average of the ratios at Screening and Day 0 Visits.

 <sup>[2]</sup> Change = Change from Baseline
 [3] One -way analysis of variance (ANOVA) with treatment group as a factor.
 [4] Nonparametric tests for differences across a one-way classification of treatment. path\t\_program.sas date time


**Protocol Number: VMCLI-II-09-002** 

ViroMed Co., Ltd.

Table 7.1.1 Ankle Brachial-Index (mmHg) – Index Leg Per-Protocol Population

| | Placebo | | VM202- 8 mg (N= ) | | | |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Desetting [1] | | | | | | |
| Baseline [1]<br>N | | | | | | |
| Mean (SD) | n<br>vv v (vv vv) | | n<br>xx.x (xx.xx) | | n<br>vv v (vv vv) | |
| Median | xx.x (xx.xx)<br>xx.x | | XX.X (XX.XX) | | xx.x (xx.xx)<br>xx.x | |
| Min, Max | XX, XX | | xx, xx | | xx, xx | |
| Day 28 | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| C : N 1 | | | | | | |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | ( ) | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| 7570 OTTOLES MEAN DIMENSIONS | | | | (AAAA, AAAA) | | (AAIA, AIAA) |
| Overall <i>p</i> -value for Treatment Differences | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Dunnett's test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. Day 28 (Paired t-test) | | x.xxxx | | x.xxxx | | x.xxxx |
| • • • | | | | | | |
| Model 2 [4] | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | X.XXXX |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Wilcoxon Rank Sum test) | | | | X.XXXX | | X.XXXX |
| Baseline vs. Day 28 (Wilcoxon Signed Rank test) | | X.XXXX | | X.XXXX | | X.XXXX |

Baseline value is the measurement taken at the Day-0 (Pre-Dose) Visit if the percent difference (= $|Day-0 - Screening|/Screening \times 100\%$ ) between the measurements taken at the Screening Visit and the Day-0 Visit is  $\leq 15\%$ . Otherwise, the baseline value is the average of the measurements taken at Screening and Day-0 Visits.

Programmer Note Repeat for all available time points, Day 28, Day 90, 6mo, 9mo and 12mo.

Programmer Note Tables 7.1.2 will be identical to Table 7.1.1 for the ITT Population using imputation rules specified in Section 10.2.3 of the Statistical Analysis Plan.

Programmer Note Tables 7.2 will be identical to Table 7.1 for the ABI – Non-Index Leg.

<sup>[2]</sup> Change = Change from Baseline

<sup>[3]</sup> One –way analysis of variance (ANOVA) with treatment group as a factor.

<sup>[4]</sup> Nonparametric tests for differences across a one-way classification of treatment. path/t program.sas date time


Protocol Number: VMCLI-II-09-002

ViroMed Co., Ltd.

**Table 8.1.1** Toe Brachial-Index (mmHg) - Index Leg **Per-Protocol Population** 

| | Placebo<br>Result | (N= )<br>Change [2] | VM202- 8<br>Result | mg (N= )<br>Change <sup>[2]</sup> | VM202- 10<br>Result | 6 mg (N= )<br>Change <sup>[2]</sup> |
|---|---|---|---|---|---|---|
| Baseline [1]<br>N | | | , | | , | |
| Mean (SD) | n<br>xx.x (xx.xx) | | n<br>xx.x (xx.xx) | | n<br>xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | |
| Day 28 | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| Overall p-value for Treatment Differences | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Dunnett's test) | | | | x.xxxx | | X.XXXX |
| Baseline vs. Day 28 (Paired t-test) | | X.XXXX | | X.XXXX | | x.xxxx |
| Model 2 [4] | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | x.xxxx |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Wilcoxon Rank Sum test) | | | | X.XXXX | | X.XXXX |
| Baseline vs. Day 28 (Wilcoxon Signed Rank test) | | X.XXXX | | X.XXXX | | X.XXXX |

Baseline value is the measurement taken at the Day-0 (Pre-Dose) Visit if the percent difference (= $|Day-0 - Screening|/Screening \times 100\%$ ) between the measurements taken at the Screening Visit and the Day-0 Visit is  $\leq 15\%$ . Otherwise, the baseline value is the average of the measurements taken at Screening and Day-0 Visits.

Programmer Note Repeat for all available time points, Day 28, Day 90, 6mo, 9mo and 12mo.

Programmer Note Tables 8.1.2 will be identical to Table 8.1.1 for the ITT Population using imputation rules specified in Section 10.2.3 of the Statistical Analysis Plan.

Programmer Note Tables 8.2 will be identical to Table 8.1 for the TBI – Non-Index Leg.

<sup>[2]</sup> Change = Change from Baseline
[3] One –way analysis of variance (ANOVA) with treatment group as a factor.

<sup>[4]</sup> Nonparametric tests for differences across a one-way classification of treatment. path\t program.sas date time


**Protocol Number: VMCLI-II-09-002** 

# **Table 9.1.1** Wound Area (cm<sup>2</sup>) **Per-Protocol Population**

| | Placebo | (N= ) | VM202- 8 | mg (N= ) | VM202- 16 | 6 mg (N= ) |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | |
| | | | | | _ | |
| N | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| Day 14 | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

 $<sup>^{[1]}</sup>$  Baseline defined as the last non-missing value prior to first dose of study drug.  $^{[2]}$  Change = Change from Baseline

Programmer Note Repeat for all available time points, Day 14, Day 28, Day 42, Day 49, Day 90, 6mo, 9mo, and 12mo. Programmer Note Tables 9.1.2 will be identical to Table 9.1.1 for the ITT Population.

path\t\_program.sas date

**Protocol Number: VMCLI-II-09-002** 

**Table 9.2.1 Categorical Analysis of Wound Healing Per-Protocol Population** 

| | Placebo<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| No Ulcers are Reported at Baseline | n (%) | n (%) | n (%) |
| 100% Healed Ulcer Post Baseline?<br>Yes | n (%) | n (%) | n (%) |
| No Overall <i>p</i> -value <sup>[1]</sup> <i>p</i> -value <i>vs</i> . Placebo <sup>[1]</sup> | n (%) | n (%)<br>x.xxxx | n (%)<br>x.xxxx<br>x.xxxx |

Programmer Note Tables 9.2.2 will be identical to Table 9.2.1 for the ITT Population.

Programmer Note Repeat for all available visit.

Note: Only subjects with ulcers at baseline are considered for analysis.

[1] p-value for treatment group difference from Fisher's exact test.

path\t\_program.sas date time


**Protocol Number: VMCLI-II-09-002** 

### **Table 10.1.1** VascuQoL - Activity Domain **Per-Protocol Population**

| | | (N= ) | VM202- 8 mg (N= ) | | | 6 mg (N= ) |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | |
| N | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| Day 90 | | | | | | |
| Ň | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| Overall p-value for Treatment Differences | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Dunnett's test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. Day 90 (Paired t-test) | | X.XXXX | | X.XXXX | | x.xxxx |
| Model 2 [4] | | | | | | |
| Overall <i>p</i> -value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Wilcoxon Rank Sum test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. Day 90 (Wilcoxon Signed Rank test) | | x.xxxx | | x.xxxx | | X.XXXX |

Note: VascuQoL Activity domain score is the total of the non-missing scores (from questions 4, 9, 10, 14, 16, 18, 22, and 24) divided by the number of responded questions in the domain.

[1] Baseline defined as the last non-missing value prior to first dose of study drug.

[2] Change = Change from Baseline

path\t\_program.sas date

Programmer Note Repeat for all available time points, 3mo, 9mo and 12mo.
Programmer Note Tables 10.1.2 will be identical to Table 10.1.1 for the ITT Population.

One –way analysis of variance (ANOVA) with treatment group as a factor.

Nonparametric tests for differences across a one-way classification of treatment.

Programmer Note Tables 10.2, 10.3, 10.4, 10.5 and 10.6 will be identical to Table 10.1 for the other domain scores (Symptom, Pain, Emotional, and Social), Total score and Resting Pain Please make change to the footnote for the score definition accordingly.

Programmer Note Table 10.7 will be identical to Table 10.1 for each individual question.

Table 11.1.1 Amputation– Event Free Probability Per-Protocol Population

| Amputation | Placebo<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| N | (0/) | ·· (0/) | ·· (0/) |
| Number (%) of Subjects Who Had Amputation | n (%) | n (%) | n (%) |
| Number (%) of Subjects Censored | n (%) | n (%) | n (%) |
| Quartiles [95% CI] (days) | | | |
| 25 <sup>th</sup> Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| 50 <sup>th</sup> Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| 75 <sup>th</sup> Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| <i>p</i> -value <sup>[1]</sup> | | x.xxxx | x.xxxx |
| Kaplan Meier Estimate (# at Risk) | | | |
| 6 Months | x.xxxx (n) | x.xxxx (n) | x.xxxx (n) |
| 12 Months | x.xxxx (n) | x.xxxx (n) | x.xxxx (n) |
| Range (days) | | | |
| Subjects with an Event | xx, xx | XX, XX | xx, xx |
| All Subjects | xx, xx | xx, xx | xx, xx |
| 3 | • | , | · |

<sup>[1]</sup> P-value tests for treatment difference using log rank test. path\t\_program.sas date time

Programmer Note Tables 11.1.2 will be identical to Table 11.1.1 for the ITT Population. Programmer Note For censoring rules, see Section 10.2.7 of the Statistical Analysis Plan.

Table 11.2.1 Limb Salvage – Event Free Probability Per-Protocol Population

| Limb Salvage | Placebo | VM202- 8 mg | VM202- 16 mg |
|---|---|---|---|
| | (N= ) | (N= ) | (N= ) |
| Number (%) of Subjects Who Had a Limb Salvage Procedure Performed Number (%) of Subjects Censored | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) |
| Quartiles [95% CI] (days) 25 <sup>th</sup> Percentile 50 <sup>th</sup> Percentile 75 <sup>th</sup> Percentile p-value [1] | xx (xx.x, xx.x)<br>xx (xx.x, xx.x)<br>xx (xx.x, xx.x) | xx (xx.x, xx.x)<br>xx (xx.x, xx.x)<br>xx (xx.x, xx.x)<br>x.xxxx | xx (xx.x, xx.x)<br>xx (xx.x, xx.x)<br>xx (xx.x, xx.x)<br>x.xxxx |
| Kaplan Meier Estimate (# at Risk)<br>6 Months<br>12 Months | x.xxxx (n)<br>x.xxxx (n) | x.xxxx (n)<br>x.xxxx (n) | x.xxxx (n)<br>x.xxxx (n) |
| Range (days) Subjects with an Event All Subjects | xx, xx | xx, xx | xx, xx |
| | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> P-value test for treatment difference using log rank test. path\t\_program.sas date time

Programmer Note Tables 11.1.2 will be identical to Table 11.1.1 for the ITT Population. Programmer Note For censoring rules, see Section 10.2.7 of the Statistical Analysis Plan.

Table 11.3.1 Mortality – Event Free Probability Per-Protocol Population

| Mortality | Placebo (N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| | ` | , , | , , |
| Number (%) of Subjects Who Expired | n (%) | n (%) | n (%) |
| Number (%) of Subjects Censored | n (%) | n (%) | n (%) |
| Quartiles [95% CI] (days) | | | |
| 25 <sup>th</sup> Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx(xx.x, xx.x) |
| 50 <sup>th</sup> Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| 75 <sup>th</sup> Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| <i>p</i> -value <sup>[1]</sup> | | X.XXXX | X.XXXX |
| Kaplan Meier Estimate (# at Risk) | | | |
| 6 Months | x.xxxx (n) | x.xxxx (n) | x.xxxx (n) |
| 12 Months | x.xxxx (n) | x.xxxx (n) | x.xxxx (n) |
| Range (days) | | | |
| Subjects with an Event | xx, xx | xx, xx | xx, xx |
| All Subjects | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> P-value test for treatment difference using log rank test. path\t\_program.sas date time

Programmer Note Tables 11.1.2 will be identical to Table 11.1.1 for the ITT Population. Programmer Note For censoring rules, see Section 10.2.7 of the Statistical Analysis Plan.

ViroMed Co., Ltd. Page x of x

Protocol Number: VMCLI-II-09-002

# **Table 12.1 Rutherford Classification of Disease Severity Per-Protocol Population**

| | Placebo | o (N= ) | VM202- 8 mg (N= ) | | VM202- 1 | 6 mg (N= ) |
|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | |
| N | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| 6 Months | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx |
| Comparison vs. Placebo | | | | | | |
| Model 1 [3] | | | | | | |
| LS Means (SE) | | xx.x (xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| LS Mean Differences (SE) | | | | xx.x (xx) | | xx.x (xx) |
| 95% CI for LS Mean Differences | | | | (xx.x, x.xx) | | (xx.x, x.xx) |
| Overall <i>p</i> -value for Treatment Differences | | | | | | x.xxxx |
| Pairwise p-value vs. Placebo (Dunnett's test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 6 Months (Paired t-test) | | X.XXXX | | X.XXXX | | x.xxxx |
| Model 2 [4] | | | | | | |
| Overall p-value for Treatment Differences (Jonckherre-Terpstra test) | | | | | | X.XXXX |
| Pairwise <i>p</i> -value <i>vs.</i> Placebo (Wilcoxon Rank Sum test) | | | | x.xxxx | | x.xxxx |
| Baseline vs. 6 Months (Wilcoxon Signed Rank test) | | X.XXXX | | X.XXXX | | X.XXXX |

Programmer Note Repeat for all available time point, 6mo, 9mo and 12mo.
Programmer Note Tables 12.2 will be identical to Table 12.1 for the ITT Population.

Baseline defined as the last non-missing value prior to first dose of study drug.

Change = Change from Baseline

One -way analysis of variance (ANOVA) with treatment group as a factor.

Nonparametric tests for differences across a one-way classification of treatment. path\t program.sas date time

Table 13
Study Drug Exposure
Safety Population

| | Placebo<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| | (14- ) | (14- ) | (14 ) |
| Day 0 | | | |
| Dose Administered? | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Zone of Injections [1] | | | |
| Ĭ | n (%) | n (%) | n (%) |
| II | n (%) | n (%) | n (%) |
| III | n (%) | n (%) | n (%) |
| IV | n (%) | n (%) | n (%) |
| Total Volume Administered per Protocol? | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Duration of Dose Administration (min) | | | |
| N | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Day 14 | | | |
| Dose Administered? | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Etc. | | | ••• |

 $<sup>^{[1]}</sup>$  Percentage may add up to more than 100% because more than 1 zone can be reported per subject. path\t\_program.sas  $\quad$  date  $\quad$  time

Programmer Note Repeat for all available time point,. Day 14, Day 28, and Day 42.

Protocol Number: VMCLI-II-09-002

Table 14
Treatment Emergent Adverse Events by System Organ Class and Preferred Term
Safety Population

| | | Placebo (N= ) VM202- 8 mg (N= ) | | | VM202- 16 | mg (N= ) |
|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Number of Subjects [1] | Number of<br>Events | Number of Subjects [1] | Number of<br>Events | Number of Subjects [1] | Number of<br>Events |
| Subjects Reporting at Least One Adverse Event | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n<br>n<br>n | n (%)<br>n (%)<br>n (%) | n<br>n<br>n | n (%)<br>n (%)<br>n (%) | n<br>n<br>n |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n<br>n<br>n | n (%)<br>n (%)<br>n (%) | n<br>n<br>n | n (%)<br>n (%)<br>n (%) | n<br>n<br>n |

Etc.

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once. path\t\_program.sas date time

Protocol Number: VMCLI-II-09-002

Table 15
Treatment Emergent Adverse Events by Maximum Severity
Safety Population

| | | Placebo (N= ) | | VM202- 8 mg (N= ) VM202- 16 mg ( | | | 1202- 16 mg (N= | ) | |
|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

Etc.

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the highest severity. path\t program.sas date time

Protocol VMCLI-II-09-002 Statistical Analysis Plan CONFIDENTIAL


Protocol Number: VMCLI-II-09-002

Table 16 Treatment Emergent Adverse Events by Relationship to Study Drug **Safety Population** 

| | | | Placebo (N= ) VM202- 8 mg (N= ) | | VM202- 16 | 1202- 16 mg (N= ) |
|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Related [1] | Unrelated [2] | Related [1] | Unrelated [2] | Related [1] | Unrelated [2] |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 Preferred Term 2 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| ·<br>· | | | | | | |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the closest relationship to study drug.

[1] Includes all events reported as "Possibly," "Probably," "Definitely" or with missing relationship to study drug.

[2] Includes all events reported as "Not Related" relationship to study drug.

path\t\_program.sas date time

**Protocol Number: VMCLI-II-09-002** 

Table 17 Treatment Emergent Serious Adverse Events by System Organ Class and Preferred Term **Safety Population** 

| | | (N= ) | VM202- 8 m | ıg (N= ) | VM202- 16 mg (N= ) | |
|---|---|---|---|---|---|---|
| | Number of | Number of | Number of | Number of | Number of | Number of |
| System Organ Class / Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Serious Adverse Event | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |
| ·<br>· | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |

Etc.

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once. path\t\_program.sas date

Protocol Number: VMCLI-II-09-002

## Table 18 Hematology - Shift from Baseline Safety Population Analyte #1

Baseline [1]

| | Placebo (N= ) | | | VM202- 8 mg (N= ) | | | VM202- 16 mg (N= ) | | = ) |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| Day 14 | | n | | | n | | | n | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 28 | | n | | | n | | | n | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Etc.

Programmer Note Analytes to be shown include Hematocrit, Hemoglobin, RBC, WBC, Platelets, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, MCV, MCHC, MCH.

<sup>[1]</sup> Baseline defined as the last non-missing value prior to first dose of study drug. path\t\_program.sas date time

Protocol Number: VMCLI-II-09-002

## Table 19 Serum Chemistry - Shift from Baseline Safety Population Analyte #1

Baseline [1]

| | Placebo (N= ) | | | VM202- 8 mg (N= ) | | | VM202- 16 mg (N= ) | | [= ) |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| Day 14 | | n | | | n | | | n | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 28 | | n | | | n | | | n | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Etc.

Programmer Note Analytes to be shown include Albumin, Alkaline Phosphate, ALT, AST, Bicarbonate, BUN, Calcium, Chloride, Creatinine, GGT Glucose, LDH, Phosphorus, Sodium, Total Bilirubin, Total Protein, Uric Acid.

<sup>[1]</sup> Baseline defined as the last non-missing value prior to first dose of study drug. path\t\_program.sas date time

Protocol Number: VMCLI-II-09-002

Table 20 Vital Signs **Safety Population** 

| | Placebo (N= ) | | VM202- 8 | mg (N= ) | VM202- 16 mg (N= ) | |
|---|---|---|---|---|---|---|
| Vital Sign | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Heart Rate (bpm) | | | | | | |
| Baseline [1] | | | | | | |
| N | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | XX, XX | |
| Day 0 (Post Dose) | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 14 (Pre- Dose) | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |
| Day 14 (Post-Dose) | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

Etc.

Programmer Note Repeat for all available time points and vital signs.

Baseline defined as the last non-missing value prior to first dose of study drug.
 Change = Change from Baseline
 path\t\_program.sas
 date
 time

**Protocol Number: VMCLI-II-09-002** 

### Table 21 Retinal Fundoscopy- Shift from Baseline **Safety Population**

Screening/Baseline ----- Placebo (N= ) ---------- VM202- 8 mg (N= ) ---------- VM202- 16 mg (N= ) -----Abn, Not Abn, Abn, Not Abn, Abn, Not Abn,  $CS^{[1]}$ CS [2]  $CS^{[1]}$ CS [2]  $CS^{[1]}$ CS [2] Normal Normal Normal 12 Months Right n (%) n (%) n (%) Normal n (%) n (%) n (%) n (%) n (%) n (%) Abnormal, Not Clinically Significant n (%) Abnormal, Clinically Significant n (%) Left n n Normal n (%) Abnormal, Not Clinically Significant n (%) Abnormal, Clinically Significant n (%)

Note: In the case of an early withdrawal, the result from the last retinal fundoscopy is considered for the 12 Months visit.

path\t program.sas date time

<sup>[1]</sup> Abn, Not CS= Abnormal, Not Clinically Significant

<sup>[2]</sup> Abn, CS= Abnormal, Clinically Significant

Table 22
Injection Site Reaction
Safety Population

| | Placebo<br>(N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| ubject reported an Injection Site Reaction? | (11 | (14 ) | (11 |
| Day 0 (Post-Dose) | n | n | n |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Day14 (Pre-Dose) | n | n | n |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Day14 (Post-Dose) | n | n | n |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Etc. | | | |
| time | | | |

path\t\_program.sas date time

Programmer Note Repeat for all available time point, Day 28(pre- and post-dose), Day 42(pre- and post-dose), and Day 49(pre- and post-dose).

Protocol Number: VMCLI-II-09-002

Table 23
Prior and Concomitant Medications
Safety Population

| ATC Drug Class / Medication Term | Placebo (N= ) | VM202- 8 mg<br>(N= ) | VM202- 16 mg<br>(N= ) |
|---|---|---|---|
| | (0/) | (0/) | (0/) |
| Subjects Receiving any Concomitant Medications | n (%) | n (%) | n (%) |
| Drug Class 1 | n (%) | n (%) | n (%) |
| Medication Term 1 | n (%) | n (%) | n (%) |
| Medication Term 2 | n (%) | n (%) | n (%) |
| • | | | |
| Drug Class 2 | n (%) | n (%) | n (%) |
| Medication Term 1 | n (%) | n (%) | n (%) |
| Medication Term 2 | n (%) | n (%) | n (%) |
| Etc. | | | |

Note: At each level of summation (overall, ATC drug class, medication term), subjects reporting more than medication are counted only once. path\t\_program.sas date time

# **APPENDIX C: FIGURE LAYOUTS**

ViroMed Co., Ltd. Protocol Number: VMCLI-II-09-002

Figure 1 Amputation– Event Free Probability Safety Population



Programmer note Figure 2 and Figure 3 will be identical to Figure 1 for Limb Salvage and Mortality Event free Probability.

APPENDIX D: LISTING LAYOUTS


Protocol Number: VMCLI-II-09-002

# Listing 1 **Subject Disposition**

| Treatment Group | Subject<br>ID | ITT Population [1] | Safety<br>Population <sup>[2]</sup> | Per-Protocol<br>Population [3] | Informed<br>Consent date<br>(Study Day) | Date of First<br>Dose<br>(Study Day) | Date of Exit<br>(Study Day) | Completed the Study? | If No, Primary Reason for Premature Discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxx | Yes/No | Yes/No | Yes/No | Date9. (x) | Date9. (x) | Date9. (x) | Yes/No | Reason |
| 1 laccoo | XXXX | Yes/No | Yes/No | Yes/No | Date 9. (x) | Date 9. (x) | Date 9. (x) | Yes/No | Reason |
| VM202- 8 mg | XXXX | Yes/No | Yes/No | Yes/No | Date9. (x) | Date9. (x) | Date9. (x) | Yes/No | Reason |
| | XXXX | Yes/No | Yes/No | Yes/No | Date9. (x) | Date9. (x) | Date9. (x) | Yes/No | Reason |
| VM202- 16 mg | XXXX | Yes/No | Yes/No | Yes/No | Date9. (x) | Date9. (x) | Date9. (x) | Yes/No | Reason |
| | XXXX | Yes/No | Yes/No | Yes/No | Date9. (x) | Date9. (x) | Date9. (x) | Yes/No | Reason |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

[1] All subjects who were randomized regardless of whether treatment was received.

[2] All subjects who received at least one dose of study drug.

[3] All subjects who received the correct dose of study drug medication, have the 9-month VAS assessment, and do not have any protocol violations or major deviations. path\t program.sas date time

Protocol Number: VMCLI-II-09-002

Listing 2
Protocol Deviations

| Treatment<br>Group | Subject<br>ID | Date of<br>Deviation<br>(Study Day) | Deviation<br>Classification | Deviation | Action Taken | IRB Notification<br>Date<br>(Study Day) |
|---|---|---|---|---|---|---|
| Placebo | xxxx | Date9. (x) | Deviation Type | Deviation Description | Inclusion/Exclusion # | Date9. (x) |
| | | Date9. (x) | Deviation Type | Deviation Description | Inclusion/Exclusion # | Date9. (x) |
| VM202-8 mg | XXXX | Date9. (x) | Deviation Type | Deviation Description | Inclusion/Exclusion # | Date9. (x) |
| | | Date9. (x) | Deviation Type | Deviation Description | Inclusion/Exclusion # | Date9. (x) |
| VM202-16 mg | XXXX | Date9. (x) | Deviation Type | Deviation Description | Inclusion/Exclusion # | Date9. (x) |
| | | Date9. (x) | Deviation Type | Deviation Description | Inclusion/Exclusion # | Date9. (x) |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer Note Data comes from external excel spreadsheet. Protocol Deviations will not be directly recorded onto CRFs.

Protocol Number: VMCLI-II-09-002

# Listing 3 Eligibility Criteria

| Treatment Group | Subject<br>ID | Met All<br>Eligibility Criteria? | Criteria Not Met | Date Waiver Granted | Exemption Explanation | Exemption Granted By |
|---|---|---|---|---|---|---|
| Placebo | xxxx | Yes/No | Inclusion/Exclusion # | Date9. | Explanation. | Name |
| 1 14000 | XXXX | Yes/No | Inclusion/Exclusion # | Date9. | Explanation. Explanation. | Name |
| | | 1 63/140 | metasion/Exclusion # | Date). | Explanation. | Name |
| VM202- 8 mg | XXXX | Yes/No | Inclusion/Exclusion # | Date9. | Explanation. | Name |
| 5 | XXXX | Yes/No | Inclusion/Exclusion # | Date9. | Explanation. | Name |
| | ••• | | | | | |
| VM202- 16 mg | XXXX | Yes/No | Inclusion/Exclusion # | Date9. | Explanation. | Name |
| | XXXX | Yes/No | Inclusion/Exclusion # | Date9. | Explanation. | Name |

path\t\_program.sas date time

**Protocol Number: VMCLI-II-09-002** 

Listing 4 **Demographics and Baseline Characteristics** 

| Treatment Group | Subject ID | Date of Birth | Age (years) <sup>[1]</sup> | Sex | Race | Weight (lb)[2] | Height (in)[3] |
|---|---|---|---|---|---|---|---|
| Placebo | Xxxx | Date9. | XX | Sex | Race | XX.X | xxx.x |
| | Xxxx | Date9. | XX | Sex | Race | XX.X | XXX.X |
| VM202- 8 mg | <br>Xxxx | Date9. | *** | Sex | Race | *** ** | ***** |
| V1V12U2- 8 IIIg | Xxxx | Date9. | XX<br>XX | Sex | Race | XX.X<br>XX.X | XXX.X<br>XXX.X |
| | | | | _ | _ | | |
| VM202- 16 mg | Xxxx | Date9. | XX | Sex | Race | XX.X | XXX.X |
| | Xxxx | Date9. | XX | Sex | Race | XX.X | XXX.X |

Age calculated by determining the number of years between the date of informed consent and the date of birth.
Result collected at Day 0. If Day 0 result not collected, then the Screening result will be displayed.
Result collected at Screening.
path\t\_program.sas date time

Protocol Number: VMCLI-II-09-002

# Listing 5 Medical History

| Treatment | Subject | Diabetes | Renal | MIL# | D - 1 C | Description | Year of | Onesine |
|---|---|---|---|---|---|---|---|---|
| Group | ID | Mellitus | Dysfunction | MH# | Body System | Description | Onset | Ongoing |
| Placebo | xxxx | Yes/No | Yes/No | 1<br>2 | Body System<br>Body System | Description Description | Year4.<br>Year4. | Yes/No<br>Yes/No |
| VM202- 8 mg | xxxx | Yes/No | Yes/No | 1<br>2 | Body System<br>Body System | Description<br>Description | Year4.<br>Year4. | Yes/No<br>Yes/No |
| VM202- 16 mg | xxxx | Yes/No | Yes/No | 1 2 | Body System<br>Body System | Description<br>Description | Year4.<br>Year4. | Yes/No<br>Yes/No |

path\t\_program.sas date time

Programmer note Listing should be sorted by MH # within a subject.

Protocol Number: VMCLI-II-09-002

Listing 6
Peripheral Vascular Disease Intervention History

| Treatment | Subject | PVDIH | Date of Intervention | | | Surgical Materials | |
|---|---|---|---|---|---|---|---|
| Group | ID | # | (Study Day) | Type | Surgical Site | Used | Leg |
| Placebo | xxxx | 1 | date9. (xx) | Description | Description | Description | left/right |
| | | 2 | date9. (xx) | Description | Description | Description | left/right |
| VM202- 8 mg | XXXX | 1 | date9. (xx) | Description | Description | Description | left/right |
| | | 2 | date9. (xx) | Description | Description | Description | left/right |
| VM202- 16 mg | XXXX | 1 | date9. (xx) | Description | Description | Description | left/right |
| | | 2 | date9. (xx) | Description | Description | Description | left/right |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note Listing should be sorted by PVDIH # within a subject.

**Protocol Number: VMCLI-II-09-002** 

# Listing 7 Physical Examination at Screening

| Treatment Group | Subject<br>ID | Visit | Date of<br>Examination<br>(Study Day) | Any Abnormal<br>Findings on the<br>Physical<br>Examination? | Body System | Description of Abnormality |
|---|---|---|---|---|---|---|
| Placebo | | Visit | date9. (xx) | Yes/No | Body system<br>Body system<br>Body system | description<br>description<br>description |
| VM202- 8 mg | | Visit | date9. (xx) | Yes/No | Body system<br>Body system<br>Body system | description<br>description<br>description |
| VM202- 16 mg | XXXXXX | Visit | date9. (xx) | Yes/No | Body system<br>Body system<br>Body system | description<br>description<br>description |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note sort by date of assessment within each subject

Programmer note Height is collected on Physical Examination page, but is reported in the Demographic and Baseline Listing.

**Protocol Number: VMCLI-II-09-002** 

### Listing 8 Chest X-Ray/CT Scan

| Treatment Group | Subject ID | Visit | Date of Scan (Study Day) | Scan Type | Result | If Abnormal, Specify: |
|---|---|---|---|---|---|---|
| Placebo | xxxxxx | Visit | date9. (xx) | x | result | |
| | xxxxxx | | date9. (xx) | X | result# | description |
| | ••• | | | | | |
| VM202- 8 mg | xxxxxx | Visit | date9. (xx) | X | result* | description |
| | xxxxxx | Visit | date9. (xx) | X | result | • |
| | ••• | | | | | |
| VM202- 16 mg | xxxxxx | Visit | date9. (xx) | X | result | |
| | xxxxxx | Visit | date9. (xx) | X | result | |
| | ••• | | | | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal - Not Clinically Significant. \* Abnormal - Clinically Significant.

path\t\_program.sas date time

Programmer note Results presented as Normal or Abnormal.

Protocol Number: VMCLI-II-09-002

# Listing 9 Infection Screening

| | | | Collection Date | | | HBcAb; | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Subject ID | Visit | (Study Day) | HIV | HBsAg | IgG and IgM | HBsAb | Anti-HCV | HTLV |
| Placebo | xxxxxx | Visit | date9. (xx) | X | result | result | result | result | result |
| | xxxxxx | Visit | date9. (xx) | X | result | result | result | result | result |
| | ••• | | | | | | | | |
| VM202- 8 mg | xxxxxx | Visit | date9. (xx) | x | result | result | result | result | result |
| | XXXXXX | Visit | date9. (xx) | X | result | result | result | result | result |
| VM202- 16 mg | xxxxxx | Visit | date9. (xx) | x | result | result | result | result | result |
| | XXXXXX | Visit | date9. (xx) | X | result | result | result | result | result |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note Results presented as Negative, Positive, or Not Done.

**Protocol Number: VMCLI-II-09-002** 

## Listing 10 Urine Pregnancy Test

| | | | Was a Urine Pregnand | Collection Date | | |
|---|---|---|---|---|---|---|
| Treatment Group | Subject ID | Visit | Test Performed? | If No, Specify Reason | (Study Day) | Result |
| Placebo | XXXXXX | Visit | Yes/No | reason | date9. (xx) | result |
| | XXXXXX | Visit | Yes/No | reason | date9. (xx) | result |
| | ••• | | | | | |
| VM202- 8 mg | xxxxxx | Visit | Yes/No | reason | date9. (xx) | result |
| C | XXXXXX | Visit | Yes/No | reason | date9. (xx) | result |
| | ••• | | | | | |
| VM202- 16 mg | xxxxxx | Visit | Yes/No | reason | date9. (xx) | result |
| C | xxxxxx | Visit | Yes/No | reason | date9. (xx) | result |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note Results presented as Negative or Positive.

**Protocol Number: VMCLI-II-09-002** 

## Listing 11 Mammogram

| Subject ID | Visit | <i>3</i> | 3 | If No, specify: | Date of<br>Mammogram<br>(Study Day) | Result | If Abnormal, Specify: |
|---|---|---|---|---|---|---|---|
| xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No<br>Yes/No | Yes/No<br>Yes/No | description<br>description | date9. (xx)<br>date9. (xx) | result<br>Result# | description |
| xxxxxx | Visit | Yes/No | Yes/No | description | date9. (xx) | Result* | description |
| | Visit | Yes/No | Yes/No | description | date9. (xx) | result | |
| xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No<br>Yes/No | Yes/No<br>Yes/No | description<br>description | date9. (xx)<br>date9. (xx) | result<br>result | |
| | XXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXX | xxxxxx Visit xxxxxx Visit xxxxxx Visit xxxxxx Visit xxxxxx Visit xxxxxx Visit xxxxxx Visit | Subject ID Visit Past 12 Months? [1] XXXXXX Visit XXXXXX Visit XYes/No XXXXXX Visit Yes/No XXXXXX Visit Yes/No XXXXXX Visit XYes/No XXXXXX Visit Yes/No XXXXXX Visit Yes/No XXXXXX Visit Yes/No XXXXXX Visit Yes/No | Mammogram in the Past 12 Months? [1] Mammogram in the Past 12 Months? [2] | Subject ID Visit Past 12 Months? [1] XXXXXX Visit Yes/No Yes/No Yes/No description XXXXXX Visit Yes/No Xes/No Xes | Subject ID Mammogram in the Past 24 Months? 19 24 Months? 19 24 Months? 19 15 No, specify: (Study Day) | Mammogram in the Past Mammogram on the Past Mammogram |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. Note: # Abnormal – Not Clinically Significant; \* Abnormal - Clinically Significant.

path\t program.sas date time

Programmer note Results presented as Normal or Abnormal.

<sup>[1]</sup> For subjects in the US.

<sup>[2]</sup> For subjects in Korea.


**Protocol Number: VMCLI-II-09-002** 

### Listing 12 **PAP Smear**

| Treatment Group | Subject ID | Visit | J | Has the Subject Had a<br>PAP Smear in the Past<br>24 Months? [2] | If No, Specify<br>Reason: | Date of PAP Smear<br>(Study Day) | Result | If Abnormal, Specify: |
|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No<br>Yes/No | Yes/No<br>Yes/No | description<br>description | date9. (xx)<br>date9. (xx) | result<br>result# | description |
| VM202- 8 mg | xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No<br>Yes/No | Yes/No<br>Yes/No | description<br>description | date9. (xx)<br>date9. (xx) | result* result | description |
| VM202- 16 mg | xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No<br>Yes/No | Yes/No<br>Yes/No | description<br>description | date9. (xx)<br>date9. (xx) | result<br>result | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. Note: # Abnormal – Not Clinically Significant; \* Abnormal - Clinically Significant.

path\t program.sas date time

Programmer note Results presented as Normal or Abnormal.

<sup>[1]</sup> For subjects in the US.

<sup>[2]</sup> For subjects in Korea.

Protocol Number: VMCLI-II-09-002

### Listing 13 12-Lead Electrocardiogram

| Treatment Group | Subject ID | Visit | Date of ECG<br>(Study Day) | Result | If Abnormal,<br>Specify: |
|---|---|---|---|---|---|
| Placebo | XXXXXX<br>XXXXXX | Visit<br>Visit | date9. (xx)<br>date9. (xx) | result<br>result* | description |
| | | | , | | 1 |
| VM202- 8 mg | XXXXXX<br>XXXXXX | Visit<br>Visit | date9. (xx)<br>date9. (xx) | result#<br>result | description |
| VM202- 16 mg | XXXXXX<br>XXXXXX | Visit<br>Visit | date9. (xx)<br>date9. (xx) | result<br>result | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. Note: # Abnormal – Not Clinically Significant; \* Abnormal - Clinically Significant.

path\t\_program.sas date time

Programmer note Results presented as Normal or Abnormal.

Programmer note If No or Not Done is recorded on the CRF to indicate that ECG measurements were not collected, show "Not Done" under the Date of ECG column.

Protocol Number: VMCLI-II-09-002

### Listing 14 Fecal Occult Blood Test

| Treatment Group | Subject ID | Visit | Has the Subject Had a Fecal<br>Occult Blood Test in the<br>Past 12 Months? | If NO, Specify: | Date of Fecal Occult<br>Blood Test<br>(Study Day) | Result | If Abnormal, Specify: |
|---|---|---|---|---|---|---|---|
| Placebo | Xxxxxx<br>Xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | description<br>description | date9. (xx)<br>date9. (xx) | result<br>result* | description |
| VM202- 8 mg | Xxxxxx<br>Xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | description<br>description | date9. (xx)<br>date9. (xx) | result#<br>result | description |
| VM202- 16 mg | Xxxxxx<br>Xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | description description | date9. (xx)<br>date9. (xx) | result<br>result | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: NA=Subject is < 50 years old. # Abnormal – Not Clinically Significant; \* Abnormal - Clinically Significant.

path\t\_program.sas date time

Programmer note Results presented as Normal or Abnormal.

Protocol Number: VMCLI-II-09-002

#### Listing 15 Gastroscopy

| Treatment Group | Subject ID | Visit | Has the Subject Had a<br>Gastroscopy in the Past 24<br>Months? | If NO, Specify: | Date of Gastroscopy<br>(Study Day) | Result | If Abnormal, Specify: |
|---|---|---|---|---|---|---|---|
| Placebo | Xxxxxx<br>Xxxxxx<br> | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | description<br>description | date9. (xx)<br>date9. (xx) | result<br>result* | description |
| VM202- 8 mg | Xxxxxx<br>Xxxxxx<br> | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | description<br>description | date9. (xx)<br>date9. (xx) | result#<br>result | description |
| VM202- 16 mg | Xxxxxx<br>Xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | description description | date9. (xx)<br>date9. (xx) | result<br>result | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: NA=Subject is < 40 years old, has a normal result of CEA (Carcinoembryonic Antigen) and CA (Cancer Antigen) 19-9 and/or does NOT have a family history of gastric cancer.

# Abnormal - Not Clinically Significant; \* Abnormal - Clinically Significant.

path\t\_program.sas date time

Programmer note Results presented as Normal or Abnormal.

Protocol Number: VMCLI-II-09-002

#### Listing 16 Colonoscopy

| Treatment Group | Subject ID | Visit | Has the Subject Had a<br>Colonoscopy in<br>the Past 10 Years? [1] | Has the Subject Had a<br>Colonoscopy in<br>the Past 12 Months? [2] | If No, Specify<br>Reason: | Date of Colonoscopy<br>(Study Day) | Result | If Abnormal, Specify: |
|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | Yes/No/NA<br>Yes/No/NA | description<br>description | date9. (xx)<br>date9. (xx) | result<br>result# | description |
| VM202- 8 mg | xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | Yes/No/NA<br>Yes/No/NA | description<br>description | date9. (xx)<br>date9. (xx) | result* result | description |
| VM202- 16 mg | xxxxxx<br>xxxxxx | Visit<br>Visit | Yes/No/NA<br>Yes/No/NA | Yes/No/NA<br>Yes/No/NA | description description | date9. (xx)<br>date9. (xx) | result<br>result | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. Note: For subjects in the US, NA=Subject is < 50 years old.

For subjects in Korea, NA=Subject is < 50 years old, has a normal result of fecal occult blood test and/or NOT have a family history of colon cancer # Abnormal – Not Clinically Significant; \* Abnormal - Clinically Significant.

path\t\_program.sas date time

Programmer note Results presented as Normal or Abnormal.

<sup>[1]</sup> For subjects in the US.

<sup>[2]</sup> For subjects in Korea.

Protocol Number: VMCLI-II-09-002

#### Listing 17 Tumor Markers

| Treatment Group | Subject ID | Visit | Collection Date<br>(Study Day) | PSA (ng/mL) | CEA (ng/mL) | AFP (ng/mL) | CA 19-9 (U/mL) | Ca 125 (U/mL) |
|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx<br>xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | | | | | xxx.x[1/2/3]/NA[4/5/6]<br>xxx.x[1/2/3]/NA[4/5/6] |
| VM202- 8 mg | xxxxxx<br>xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | | | | | xxx.x[1/2/3]/NA[4/5/6]<br>xxx.x[1/2/3]/NA[4/5/6] |
| VM202- 16 mg | xxxxxx<br>xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | | | | | xxx.x[1/2/3]/NA[4/5/6]<br>xxx.x[1/2/3]/NA[4/5/6] |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: PSA=Prostate Specific Antigen; CEA=Carcinoembryonic Antigen; AFP=Alpha Fetoprotein; CA=Cancer Antigen. [1] Normal.

Note: Codes for Numeric Results-[1]= Normal;[2] Abnormal-Not Clinically Significant.; [3] Abnormal - Clinically Significant.

Note: Codes for NA Results- [4] Subject is female - for subject in the US and Korea.;[5] Subject is < 40 years old - for subject in Korea only.;[6] Subject is male - for subject in Korea only.

path\t program.sas date time

Programmer note Results presented as Negative, Positive, or Not Done.

Protocol Number: VMCLI-II-09-002

## Listing 18 Visual Analog Scale (VAS) for Pain

| Treatment Group | Subject ID | Visit | Assessment Date (Study Day) | Reader 1 Score<br>(mm) | Reader 2 Score (mm) | Comments |
|---|---|---|---|---|---|---|
| · | - | | | | | |
| Placebo | xxxxxx | Visit | date9. (xx) | XXX | XXX | description |
| | XXXXXX | Visit | date9. (xx) | XXX | XXX | description |
| VM202- 8 mg | XXXXXX | Visit | date9. (xx) | XXX | XXX | description |
| | XXXXXX | Visit | date9. (xx) | XXX | XXX | description |
| | ••• | | | | | |
| VM202- 16 mg | xxxxxx | Visit | date9. (xx) | xxx | xxx | description |
| V 1V1202- 10 mg | | | ` / | | | |
| | XXXXXX | Visit | date9. (xx) | XXX | XXX | description |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note sort by assessment date within each subject.

Protocol Number: VMCLI-II-09-002

# Listing 19 Resting Transcutaneous Oxygen Pressure (TcPO 2) Measurements

| Treatment<br>Group | Subject ID | Visit | Date of Assessment<br>(Study Day) | Anterior Chest<br>(mmHg) | Dorsal Surface of Foot (mmHg) | Anterior Surface of Calf (mmHg) | Posterior Surface of<br>Calf (mmHg) | Comments |
|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | result<br>result | result/Not Done result/Not Done | result/Not Done result/Not Done | result/Not Done<br>result/Not Done | comments comments |
| VM202- 8 mg | <br>xxxxxx | Visit<br>Visit | date9. (xx) date9. (xx) | result<br>result | result/Not Done<br>result/Not Done | result/Not Done<br>result/Not Done | result/Not Done<br>result/Not Done | comments comments |
| VM202- 16 mg | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | result<br>result | result/Not Done<br>result/Not Done | result/Not Done<br>result/Not Done | result/Not Done<br>result/Not Done | comments comments |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note sort by date of assessment within each subject

Programmer note If No or Not Done is recorded on the CRF to indicate that TcPO2 measurements were not collected, show "Not Done" under the Date of Assessment column.

Protocol Number: VMCLI-II-09-002

# Listing 20 Resting Ankle Brachial Index (ABI) Measurements

| | | | | Brachial<br>Press | 2 | Ankle Systolic Pressure - Right | | Ankle Systolic Pressure - Left | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>ID | Visit | Date of<br>Assessment<br>(Study Day) | Right/Left | Highest<br>Average<br>Pressure<br>(mmHg) | Pressure | PT<br>Average<br>Pressure<br>(mmHg) | (mmHg) | Resting<br>ABI | Could not<br>be<br>g Determined,<br>Explain: | Pressure | Pressure | Highest<br>Average<br>Pressure<br>(mmHg)<br>[DP/PT] [1] | | Could not be<br>Determined,<br>Explain: | Comments |
| Placebo | xxxxxx<br> | Visit<br>Visit | Date9. (xx)<br>Date9. (xx) | right/left<br>right/left | XXX.X<br>XXX.X | xxx.x<br>xxx.x | | xxx.x[x]<br>xxx.x[x] | x.xx | xxxxxx | xxx.x<br>xxx.x | | xxx.x[x]<br>xxx.x[x] | x.xx | xxxxxx | |
| VM202- 8 mg | xxxxxx<br> | Visit<br>Visit | Date9. (xx) Date9. (xx) | right/left<br>right/left | xxx.x<br>xxx.x | xxx.x<br>xxx.x | XXX.X<br>XXX.X | xxx.x[x]<br>xxx.x[x] | x.xx | xxxxxx | xxx.x<br>xxx.x | XXX.X<br>XXX.X | xxx.x[x]<br>xxx.x[x] | x.xx | xxxxxx | |
| VM202- 16 mg | | Visit<br>Visit | Date9. (xx) Date9. (xx) | right/left<br>right/left | XXX.X<br>XXX.X | xxx.x<br>xxx.x | | xxx.x[x]<br>xxx.x[x] | x.xx<br>x.xx | | xxx.x<br>xxx.x | | xxx.x[x]<br>xxx.x[x] | x.xx<br>x.xx | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.  $^{[1]}$  1=DP, 2=PT.

path\t\_program.sas date time

Programmer note sort by date of assessment within each subject Programmer note listing may need to be split over 2 pages.

Protocol Number: VMCLI-II-09-002

# Listing 21 Resting Toe Brachial Index (TBI) Measurements

| | | | | | Brachial Systo | lic Pressure | Toe Pressure - Right | | Toe Pressure - Left | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>ID | Visit | Date of<br>Assessment<br>(Study Day) | Type of<br>Equipment Used | Right/Left | Highest<br>Average<br>Pressure<br>(mmHg) | Average<br>(mmHg) | TBI | Could not be<br>Determined, Explain: | Average<br>(mmHg) | TBI | Could not be<br>Determined, Explain: | Comments |
| Placebo | xxxxxx | Visit<br>Visit | Date9. (xx) Date9. (xx) | PPG/Doppler<br>PPG/Doppler | right/left<br>right/left | xxx.x<br>xxx.x | xxx.x<br>xxx.x | x.xx | xxxxxx | XXX.X<br>XXX.X | x.xx | xxxxxx | |
| VM202- 8 mg | xxxxxx | Visit<br>Visit | Date9. (xx)<br>Date9. (xx) | PPG/Doppler<br>PPG/Doppler | right/left<br>right/left | XXX.X<br>XXX.X | XXX.X<br>XXX.X | x.xx<br>x.xx | | XXX.X<br>XXX.X | x.xx<br>x.xx | | |
| VM202- 16 mg | xxxxxx | Visit<br>Visit | Date9. (xx)<br>Date9. (xx) | PPG/Doppler<br>PPG/Doppler | right/left<br>right/left | XXX.X<br>XXX.X | XXX.X<br>XXX.X | x.xx<br>x.xx | | xxx.x<br>xxx.x | x.xx<br>x.xx | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note sort by date of assessment within each subject Programmer note listing may need to be split over 2 pages.

...

Protocol Number: VMCLI-II-09-002

ViroMed Co., Ltd.

Listing 22
Ulcer and Wound Assessment / Skin Condition Assessment

| | | | Assessment Date | Does the Subject Have<br>Ulcers Present/Same | Does the Subject Have<br>New Ulcers NOT Present at | | Skin Condition Ass | essment |
|---|---|---|---|---|---|---|---|---|
| Treatment Group | Subject ID | Visit | (Study Day) | Ulcer Still Existing? | Screening/Day 0? | Not Done | Scaling | Erythema |
| Placebo | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | Yes/No<br>Yes/No | | result<br>result | result<br>result |
| VM202- 8 mg | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | Yes/No<br>Yes/No | | result<br>result | result<br>result |
| | | | ••• | | | | | |
| VM202- 16 mg | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | Yes/No<br>Yes/No | Not Done | result | result |
| | | | ••• | | | | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. Note: 0 = No Scaling/Erythema, 1 = Very Slight, 2 = Well-defined, 3 = Moderate to Severe, 4 = Sever. path\t\_program.sas date time

Programmer note sort by date of assessment within each subject

Protocol Number: VMCLI-II-09-002

### Listing 23 Ulcer Assessment

Ulcer Status

| Treatment Group | Subject ID | Anatomical<br>Location <sup>[1]</sup> | Visit Date<br>(Study Day) | Visit | Photo and Tracings Submitted to CPC | 100% Healed | Comments |
|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx<br> | 1or 2 | date9. (xx)<br>date9. (xx) | Screen<br>Day 0 | result<br>result | result<br>result | comment |
| VM202- 8 mg | xxxxxx<br> | 1or 2 | date9. (xx)<br>date9. (xx) | Screen<br>Day 0 | result<br>result | result<br>result | comment<br>comment |
| VM202- 16 mg | xxxxxx | 1or 2 | date9. (xx)<br>date9. (xx) | Screen<br>Day 0 | result<br>result | result<br>result | comment<br>comment |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. 1 = Vascular, 2 = Non-Vascular.

path\t\_program.sas date time

Programmer note sort by time point within each subject.

Time points include Screen, Day 0, Day 14, Day 28, Day 42, Day 49, Day 90, 6 Month, 9 Month, 12 Month, USV #1, USV #2, USV #3, Early Exit.

Protocol Number: VMCLI-II-09-002

### Listing 24 Vascular Quality of Life (VascuQoL) Part 1 of 2

| Treatment Group | Subject ID | Visit | Was the VascuQoL<br>Completed this Visit? | If Yes, Assessment Date<br>(Study Day) | If No, Specify Reason: |
|---|---|---|---|---|---|
| Placebo | xxxxxx | Visit | Yes/No | date9. (xx) | description |
| 1 | XXXXXX | Visit | Yes/No | date9. (xx) | description |
| VM202- 8 mg | xxxxxx | Visit | Yes/No | date9. (xx) | description |
| | xxxxxx | Visit | Yes/No | date9. (xx) | description |
| | ••• | | | | |
| VM202- 16 mg | xxxxxx | Visit | Yes/No | date9. (xx) | description |
| • | XXXXXX | Visit | Yes/No | date9. (xx) | description |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t program.sas date time

Programmer note sort by assessment date within each subject.

Protocol Number: VMCLI-II-09-002

#### Listing 24 Vascular Quality of Life (VascuQoL) Part 2 of 2

| | | | Assessment<br>Date | Question | | | |
|---|---|---|---|---|---|---|---|
| Treatment Group | Subject ID | Visit | (Study Day) | Number | | Question Answer | Score [1] |
| Placebo | xxxxxx | Visit | date9. (xx) | 1 | During the past two weeks, I have had pain in my leg (or foot) when walking | description | 1-7 |
| | | | | 2 | During the past two weeks, I have been worried that I might injure my leg | description | 1-7 |
| | | | | | <del></del> | | |
| VM202- 8 mg | xxxxxx | Visit | date9. (xx) | 1 | During the past two weeks, I have had pain in my leg (or foot) when walking | description | 1-7 |
| | | | | 2 | During the past two weeks, I have been worried that I might injure my leg | description | 1-7 |
| VM202- 16 mg | xxxxxx | Visit | date9. (xx) | 1 | During the past two weeks, I have had pain in my leg (or foot) when walking | description | 1-7 |
| | | | | 2 | During the past two weeks, I have been worried that I might injure my leg | description | 1-7 |
| | | | | ••• | | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

[1] Each question is scored on a scale from 1 to 7, with 1 indicating poor quality of life and 7 indication maximum health.

path/t program.sas date time

Programmer note sort by assessment date within each subject.

Protocol Number: VMCLI-II-09-002

# Listing 25 High Resolution Magnetic Resonance Angiography (MRA)

| Treatment Group | Subject ID | Visit | Was a High Resolution MRA<br>Performed? | If Yes, Date Obtained<br>(Study Day) | If No, Explain: |
|---|---|---|---|---|---|
| Placebo | xxxxxx | Visit | Yes/No/NA<br>Yes/No/NA<br> | date9. (xx)<br>date9. (xx) | description<br>description |
| VM202- 8 mg | xxxxxx | Visit | Yes/No/NA<br>Yes/No/NA<br> | date9. (xx)<br>date9. (xx) | description<br>description |
| VM202- 16 mg | xxxxxx | Visit | Yes/No/NA<br>Yes/No/NA | date9. (xx)<br>date9. (xx) | description<br>description |
| | ••• | | ••• | | |

Note: Study  $Day = [(Date\ of\ Event)\ - (Treatment\ Start\ Date)];\ 1$  is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start\ Date'. NA=MRA not performed at this site.

path\t\_program.sas date time

Programmer note sort by assessment date within each subject.

Protocol Number: VMCLI-II-09-002

#### Listing 26 Rutherford Classification

| | | | Date of Assessment | t | |
|---|---|---|---|---|---|
| Treatment Group | Subject ID | Visit | (Study Day) | Rutherford Classification | Comments |
| Placebo | XXXXXX | visit | date9. (xx) | | comments |
| | | visit | date9. (xx) | X | comments |
| VM202- 8 mg | xxxxxx | visit | date9. (xx) | X | comments |
| | | visit | date9. (xx) | X | comments |
| VM202- 16 mg | xxxxxx | visit | date9. (xx) | X | comments |
| | | visit | date9. (xx) | X | comments |
| | | | ••• | | |

Note: Scale for Rutherford Classification-

- 0= Asymptomatic No hemodynamically
- 1= Mild Claudication
- 2= Moderate Claudication
- 3= Severe Claudication
- 4= Ischemic Rest Pain
- 5= Minor Tissue Loss Non-healing ulcer, focal gangrene with diffuse pedal ischemia
- 6= Major Tissue Loss Extending above the TM level, functional foot no longer salvageable

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

path\t program.sas date time

Programmer note sort by date of assessment within each subject

**Protocol Number: VMCLI-II-09-002** 

# Listing 27 Study Drug Administration

| | | | | | | | | | If | No, | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Start Time | Stop Time | Was Total | Reason Total | Total Volume | _ |
| Treatment | Subject | Visit Date | Was a Dose | Study Leg | | of First | of Last | Volume (8mL) | Volume Not | Administered | Injection |
| Group | IĎ | (Study Day) | Administered? | Assignment | Kit # | Injection | Injection | Administered? | Administered | (mL) | Zones |
| Placebo | XXXX | Date9. | Yes/No | left/right | XXXX | time5. | time5. | Yes/No | XXXXXXX | XX | I/II/II/IV |
| | XXXX | Date9. | Yes/No | left/right | XXXX | time5. | time5. | Yes/No | XXXXXXX | XX | I/II/II/IV |
| VM202- 8 mg | XXXX | Date9. | Yes/No | left/right | XXXX | time5. | time5. | Yes/No | XXXXXXX | XX | I/II/II/IV |
| | XXXX | Date9. | Yes/No | left/right | XXXX | time5. | time5. | Yes/No | XXXXXXX | XX | I/II/II/IV |
| VM202- 16 mg | XXXX | Date9. | Yes/No | left/right | XXXX | time5. | time5. | Yes/No | XXXXXXX | XX | I/II/II/IV |
| | XXXX | Date9. | Yes/No | left/right | XXXX | time5. | time5. | Yes/No | XXXXXXX | XX | I/II/II/IV |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t program.sas date time

Programmer note sort by visit date within each subject

**Protocol Number: VMCLI-II-09-002** 

## Listing 28 Adverse Events

| Treatment<br>Group | Subject ID | AE<br># | Adverse Event//<br>Preferred Term | Start Date<br>(Study Day) | End Date<br>(Study Day) | Severity | Treatment | Study<br>Drug<br>Action | Relationship<br>To Study<br>Drug | Relationship<br>To<br>Procedure | Relationship<br>To Underlying<br>Disease | Outcome | Serious? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxx | 1 | Adverse Event//<br>Preferred Term | Date9. | Date9. | Severity | Treatment | SDA | Relationship | Relationship | Relationship | Outcome | Yes/No |
| VM202- 8 mg | xxxx | 1 | Adverse Event//<br>Preferred Term | Date9. | Date9. | Severity | Treatment | SDA | Relationship | Relationship | Relationship | Outcome | Yes/No |
| VM202- 16 mg | xxxx | 1 | Adverse Event//<br>Preferred Term | Date9. | Date9. | Severity | Treatment | SDA | Relationship | Relationship | Relationship | Outcome | Yes/No |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note for each subject, sort by AE #

Protocol Number: VMCLI-II-09-002

### Listing 29 Serious Adverse Events

| Treatment Group | Subject ID | AE<br># | Adverse Event//<br>Preferred Term | Start Date<br>(Study Day) | End Date<br>(Study Day) | Severity | Treatment | Study<br>Drug<br>Action | Relationship<br>To Study<br>Drug | Relationship<br>To<br>Procedure | Relationship<br>To Underlying<br>Disease | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxx | 1 | Adverse Event//<br>Preferred Term | Date9. | Date9. | Severity | Treatment | SDA | Relationship | Relationship | Relationship | Outcome |
| VM202- 8 mg | xxxx | 1 | Adverse Event//<br>Preferred Term | Date9. | Date9. | Severity | Treatment | SDA | Relationship | Relationship | Relationship | Outcome |
| VM202- 16 mg | xxxx | 1 | Adverse Event//<br>Preferred Term | Date9. | Date9. | Severity | Treatment | SDA | Relationship | Relationship | Relationship | Outcome |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note for each subject, sort by AE #

ViroMed Co., Ltd.


Protocol Number: VMCLI-II-09-002

#### Listing 30 Hematology Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Collection Date<br>(Study Day) | WBC<br>(10 <sup>9</sup> /L) | Neutrophils (%) | Lymphocytes (%) | Monocytes (%) | Eosinophils (%) | Basophils (%) |
|---|---|---|---|---|---|---|---|---|---|
| - | | | \ | | | | | | |
| Placebo | xxxxxx | visit | date9. (xx) | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | visit | date9. (xx) | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | ••• | | | | | | |
| | ••• | | | | | | | | |
| VM202- 8 mg | XXXXXX | visit | date9. (xx) | xx.xx# | XX.X | xx.x | xx.x | xx.x | xx.x |
| Č | | visit | date9. (xx) | xx.xx* | XX.X | XX.X | xx.x | XX.X | XX.X |
| | ••• | | | | | | | | |
| VM202- 16 mg | xxxxxx | visit | date9. (xx) | XX.XX | xx.x | xx.x | xx.x | xx.x | xx.x |
| 7111202 TO ING | | visit | date9. (xx) | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | ••• | | | | | | | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal - Not Clinically Significant; as reported by the investigator . \* Abnormal - Clinically Significant; as reported by the investigator.

Note: H= Result above normal range; L= Result below normal range.

RBC=Red Blood Cells. WBC=White Blood Cells.

path\t\_program.sas date time

Programmer note sort by collection date within each subject.

ViroMed Co., Ltd.
Protocol Number: VMCLI-II-09-002

#### Listing 30 Hematology Part 2 of 2

| Treatment Group | Subject<br>ID | Visit | Collection Date<br>(Study Day) | Platelets (10 <sup>9</sup> /L) | RBC<br>(10 <sup>12</sup> /L) | Hemoglobin (g/dL) | Hematocrit (%) | MCHC<br>(g/dL) | MCH<br>(pg) | MCV<br>(fL) |
|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx | visit | date9. (xx) | vv v | VV VV | VV V | VV V | vv v | VV V | vv v |
| 1 laccoo | AAAAAA | visit | date9. (xx) | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| | ••• | | | | | | | | | |
| VM202- 8 mg | xxxxxx | visit | date9. (xx) | XX.X | xx.xx | xx.x | xx.x | xx.x | xx.x | XX.X |
| | | visit | date9. (xx) | XX.X | xx.xx | XX.X | XX.X | XX.X | xx.x | XX.X |
| | | | *** | | | | | | | |
| VM202-16 mg | xxxxxx | visit | date9. (xx) | XX.X | xx.xx# | xx.x | XX.X | XX.X | xx.x | xx.x |
| Č | | visit | date9. (xx) | XX.X | xx.xx* | XX.X | XX.X | XX.X | xx.x | XX.X |
| | | | ••• | | | | | | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal - Not Clinically Significant; as reported by the investigator . \* Abnormal - Clinically Significant; as reported by the investigator.

Note: H= Result above normal range; L= Result below normal range.

RBC=Red Blood Cells. WBC=White Blood Cells.

path\t\_program.sas date time

Programmer note sort by collection date within each subject

Protocol Number: VMCLI-II-09-002

#### Listing 31 Serum Chemistry Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Collection Date<br>(Study Day) | Albumin<br>(g/dL) | ALT<br>(U/L) | AST<br>(U/L) | ALK<br>(U/L) | Total Biliburin<br>(mg/dL) | LDH<br>(U/L) | GGT<br>(U/L) | Total Protein<br>(g/dL) | Bicarbonate (mEq/L) | Glucose<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx | visit<br>visit | date9. (xx)<br>date9. (xx) | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | xx.x<br>xx.x | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| VM202- 8 mg | xxxxxx | visit<br>visit | date9. (xx)<br>date9. (xx) | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| VM202- 16 mg | XXXXXX | visit<br>visit | date9. (xx)<br>date9. (xx) | xx.x<br>xx.x | XX.X<br>XX.X | xx.x<br>xx.x | XX.X<br>XX.X | xx.x<br>xx.x | XX.X<br>XX.X | XX.X<br>XX.X | xx.x<br>xx.x | xx.x<br>xx.x | xx.x<br>xx.x |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal - Not Clinically Significant; as reported by the investigator . \* Abnormal - Clinically Significant; as reported by the investigator.

Note: H= Result above normal range; L= Result below normal range.

 $ALT = alanine\ aminotransferase;\ AST = aspartate\ aminotransferase;\ ALK = alkaline\ phosphatase;\ LDH = lactate\ dehydrogenase;\ GGT = gamma-glutamyl\ transferase.\ BUN = blood\ urea\ nitrogen.$ 

path\t\_program.sas date time

Programmer note sort by collection date within each subject

Protocol Number: VMCLI-II-09-002

#### Listing 31 Serum Chemistry Part 2 of 2

| Treatment Group | Subject<br>ID | Visit | Collection Date<br>(Study Day) | Sodium<br>(mEq/L) | Potassium<br>(mEq/L) | Chloride (mmol/) | Calcium<br>(m/dL) | Phosphorus (m/dL) | BUN<br>(mg/dL) | Creatinine (mg/dL) | Uric Acid<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| DI 1 | | , | 1.0() | | | | | | | | |
| Placebo | XXXXXX | visit | date9. (xx) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | visit | date9. (xx) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | ••• | | | | | | | | |
| | ••• | | | | | | | | | | |
| VM202- 8 mg | xxxxxx | visit | date9. (xx) | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| v 1v1202- 6 mg | ΛΛΛΛΛΛ | | ` / | | | | | | | | |
| | | visit | date9. (xx) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | ••• | | | | | | | | |
| | ••• | | | | | | | | | | |
| VIM202 16 | | :-:4 | 1-4-0 () | | | | | | | | |
| VM202- 16 mg | XXXXXX | visit | date9. (xx) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | visit | date9. (xx) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | ••• | | | | | | | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal - Not Clinically Significant; as reported by the investigator . \* Abnormal - Clinically Significant; as reported by the investigator.

Note: H= Result above normal range; L= Result below normal range.

ALT = alanine aminotransferase; AST = aspartate aminotransferase; ALK = alkaline phosphatase; LDH = lactate dehydrogenase; GGT = gamma-glutamyl transferase. BUN = blood urea nitrogen.

path\t program.sas date time

Programmer note sort by collection date within each subject

Protocol Number: VMCLI-II-09-002

Listing 32 Urinalysis Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Collection Date<br>(Study Day) | Specific<br>Gravity | pН | Protein | Glucose | Ketone | Bilirubin | Blood | Nitrite | Leukocyte | Urobilinogen |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | XX.XXX<br>XX.XXX | XX.X<br>XX.X | Result#<br>Result* | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result |
| VM202- 8 mg | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | xx.xxx#<br>xx.xxx* | XX.X<br>XX.X | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result |
| VM202- 16 mg | xxxxxx | Visit<br>Visit | date9. (xx)<br>date9. (xx) | XX.XXX<br>XX.XXX | xx.x<br>xx.x | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result | result<br>result |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. Note: H= Result above normal range; L= Result below normal range. High/Low flags are only assigned to analytes with numeric results.

path\t\_program.sas date time

Programmer note sort by collection date within each subject

Protocol Number: VMCLI-II-09-002

Listing 32 Urinalysis Part 2 of 2

| Treatment Group | Subject<br>ID | Visit | Collection Date<br>(Study Day) | Was Microscopic Exam Performed? | RBC<br>(/hpf) | WBC<br>(/hpf) | Casts<br>(/hpf) |
|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx | visit<br>visit | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | result<br>result | result#<br>result* | result<br>result |
| | | | ••• | | | | |
| VM202- 8 mg | xxxxxx | visit<br>visit | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | result<br>result | result<br>result | result<br>result |
| VM202- 16 mg | xxxxxx | visit<br>visit | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | result<br>result | result<br>result | result<br>result |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal – Not Clinically Significant; as reported by the investigator. \* Abnormal - Clinically Significant as reported by the investigator.

path/t\_program.sas date time

Programmer note sort by collection date within each subject

Protocol Number: VMCLI-II-09-002

### Listing 33 Vital Signs

| Treatment Group | Subject II | O Visit/Time Point | Visit Date<br>(Study Day) | Time of Measurement | Vital Signs Collected? | Weight (lb) | Blood Pressure<br>(mmHg) | Temperature (F) | Respiration Rate (breaths/min) | Heart Rate (beats/min) |
|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxxxx<br> | Screening<br>Day xx<br>Day xx/ Pre Drug | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | Time5.<br>Time5. | xxx.x | systolic/diastolic<br>systolic/diastolic | XXX.X<br>XXX.X | xxx<br>xxx | XXX<br>XXX |
| VM202- 8 mg | xxxxxx<br> | Screening<br>Day xx<br>Day xx/ Pre Drug | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | Time5.<br>Time5. | XXX.X | systolic/diastolic<br>systolic/diastolic | XXX.X<br>XXX.X | xxx<br>xxx | xxx<br>xxx |
| VM202- 16 mg | xxxxxx<br> | Screening<br>Day xx<br>Day xx/ Pre Drug | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | Time5.<br>Time5. | XXX.X | systolic/diastolic<br>systolic/diastolic | XXX.X<br>XXX.X | xxx<br>xxx | xxx<br>xxx |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note sort by visit date within each subject

Programmer note If No or Not Done is recorded on the CRF to indicate that vital signs were not collected, show "Not Done" under the Visit Date column.

Protocol Number: VMCLI-II-09-002

# Listing 34 Copies of VM202 in Whole Blood

| Treatment Group | Subject ID | Visit | Pre/Post<br>Injection | Visit Date<br>(Study Day) | Was a Sample to Test VM202 Obtained? [1] | Time Obtained |
|---|---|---|---|---|---|---|
| Placebo | xxxxxx | visit | Pre/Post | date9. (xx) | Yes/No | Time5. |
| 1 laccoo | λλλλλλ | visit | Pre/Post | date9. (xx) | Yes/No | Time5. |
| | | | | ••• | | |
| | ••• | | | | | |
| VM202- 8 mg | xxxxxx | visit | Pre/Post | date9. (xx) | Yes/No | Time5. |
| | | visit | Pre/Post | date9. (xx) | Yes/No | Time5. |
| | | | | ••• | | |
| | ••• | | | | | |
| VM202- 16 mg | xxxxxx | visit | Pre/Post | date9. (xx) | Yes/No | Time5. |
| | | visit | Pre/Post | date9. (xx) | Yes/No | Time5. |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

[1] For Post Injection time points, result shown is to the question "Was a sample to test VM202 obtained (required between 1-3 hours post injection)?"

path\t\_program.sas date time

Programmer note sort by visit date within each subject

Protocol Number: VMCLI-II-09-002

Listing 35 Serum Hepatocyte Growth Factor (HGF)

| Treatment Group | Subject ID | Visit | Visit Date<br>(Study Day) | Was a Sample to Test<br>Serum HGF Obtained? | Time Obtained |
|---|---|---|---|---|---|
| Placebo | xxxxxx | visit | date9. (xx) | Yes/No | Time5. |
| 1 lacebo | AAAAA | visit | date9. (xx) | Yes/No | Time5. |
| | | | ••• | | |
| | ••• | | | | |
| VM202- 8 mg | xxxxxx | visit | date9. (xx) | Yes/No | Time5. |
| | | visit | date9. (xx) | Yes/No | Time5. |
| | | | ••• | | |
| | ••• | | | | |
| VM202- 16 mg | xxxxxx | visit | date9. (xx) | Yes/No | Time5. |
| Č | | visit | date9. (xx) | Yes/No | Time5. |
| | | | ••• | | |

Programmer note sort by visit date within each subject

Protocol Number: VMCLI-II-09-002


# Listing 36 Eye Examination - Retinal Fundoscopy

| Examination |
|-------------|

| | | | | (Stud | dy Day) | | Res | sults | |
|---|---|---|---|---|---|---|---|---|---|
| | Subject | | Examination | Retinal | Fluorescein | • | | | |
| Treatment Group | ID | Visit | Performed? | Fundoscopy | Angiography | OD (Right) | If Abnormal, describe: | OS(Left) | If Abnormal, describe: |
| Placebo | xxxxxx | Visit<br>Visit | Yes/No<br>Yes/No | Date9. (xx)<br>Date9. (xx) | Date9. (xx)<br>Date9. (xx) | Result<br>Result# | xxxxxxx | Result<br>Result* | xxxxxxx |
| VM202- 8 mg | xxxxxx | Visit | Yes/No | Date9. (xx) | Date9. (xx) | Result | | Result | |
| | | Visit | Yes/No | Date9. (xx) | Date9. (xx) | Result | | Result | |
| | ••• | | | | | | | | |
| VM202- 16 mg | xxxxxx | Visit | Yes/No | Date9. (xx) | Date9. (xx) | Result | | Result | |
| | | Visit | Yes/No | Date9. (xx) | Date9. (xx) | Result | | Result | |

. . .

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

Note: # Abnormal – Not Clinically Significant. \* Abnormal - Clinically Significant.

path\t\_program.sas date time

Programmer note sort by date of exam within each subject (sort by variable OSDT1). Results presented as Normal or Abnormal.

Protocol Number: VMCLI-II-09-002

# Listing 37 Injection Site Reaction

| Treatment Group | Subject ID | Visit | Pre/Post<br>Injection | Visit Date<br>(Study Day) | Was There an Injection Site<br>Reaction? [1] | If YES,<br>AE # |
|---|---|---|---|---|---|---|
| Placebo | xxxxxx | visit<br>visit | Pre/Post<br>Pre/Post | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | x<br>x |
| | | | | ` | | |
| VM202-8 mg | xxxxxx | visit<br>visit | Pre/Post<br>Pre/Post | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | x<br>x |
| VM202- 16 mg | xxxxxx | visit<br>visit | Pre/Post<br>Pre/Post | date9. (xx)<br>date9. (xx) | Yes/No<br>Yes/No | X<br>X |
| | | | | ••• | | |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'.

[1] For Pre Injection time Points, response shown is to the question "If an injection site reaction occurred at the previous visit, is it still present?"

path/t\_program.sas date time

Programmer note sort by visit date within each subject

**Protocol Number: VMCLI-II-09-002** 

### Listing 38 **Prior and Concomitant Medications**

| Treatment<br>Group | Subject<br>ID | CM# | Medication//<br>Drug Name | Start Date<br>(Study Day) | Stop Date<br>(Study Day) | Dose | Units | Route | Regimen | Indication |
|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | xxxx | 1 | Medication/Drug<br>Name | Date9.(xx) | Date9.(xx) | xxxx | unit | route | regimen | Medical History #/<br>Adverse Event #/ |
| | | 2 | Medication/Drug<br>Name | Date9.(xx) | Ongoing | xxxx | unit | route | regimen | Other: specify Medical History #/ Adverse Event #/ Other: specify |
| VM202- 8 mg | xxxx | 1 | Medication/Drug<br>Name | Date9.(xx) | Date9.(xx) | xxxx | unit | route | regimen | Medical History #/ Adverse Event #/ Other: specify |
| | | 2 | Medication/Drug<br>Name | Date9.(xx) | Ongoing | XXXX | unit | route | regimen | Medical History #/ Adverse Event #/ Other: specify |
| VM202- 16 mg | xxxx | 1 | Medication/Drug<br>Name | Date9.(xx) | Date9.(xx) | xxxx | unit | route | regimen | Medical History #/ Adverse Event #/ Other: specify |
| | | 2 | Medication/Drug<br>Name | Date9.(xx) | Date9.(xx) | xxxx | unit | route | regimen | Medical History #/ Adverse Event #/ Other: specify |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

 $\label{lem:continuous} Programmer\ Note\ \ sort\ by\ CM\ \#.$   $Programmer\ Note\ \ If\ Ongoing\ is\ marked,\ then\ show\ "Ongoing"\ in\ the\ Stop\ Date\ column.$ 

Protocol Number: VMCLI-II-09-002

# Listing 39 Prior and Concomitant Procedures

| | | | | | For Procedures Related to Peripheral Vascular Disease | |
|---|---|---|---|---|---|---|
| Treatment Group Subject | Subject ID | Procedure # | Procedure Name | Date of Procedure (Study Day) | Surgical Site | Leg |
| Placebo | xxxx | 1 | xxxx unit | date9. (xx) | description | left/right |
| | | 2 | xxxx unit | date9. (xx) | description | left/right |
| VD 4202 0 | ••• | 1 | •, | 1 ( 0 ( ) | 4 2 2 | 1.0/:14 |
| VM202- 8 mg | XXXX | 1 | xxxx unit | date9. (xx) | description | left/right |
| | | 2 | xxxx unit | date9. (xx) | description | left/right |
| VM202- 16 mg | XXXX | 1 | xxxx unit | date9. (xx) | description | left/right |
| | | 2 | xxxx unit | date9. (xx) | description | left/right |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t program.sas date time

Programmer note sort by date of procedure within each subject

Protocol Number: VMCLI-II-09-002

## Listing 40 Death Report

| Treatment Group | Subject ID | Date of Death (Study Day) | Cause of Death | Comments |
|---|---|---|---|---|
| Placebo | XXXX | Date9. (Study Day) | Description | Yes/No |
| Tideeoo | XXXX | Date9. (Study Day) | Description | Yes/No |
| | ••• | | | |
| VM202- 8 mg | XXXX | Date9. (Study Day) | Description | Yes/No |
| | XXXX | Date9. (Study Day) | Description | Yes/No |
| | ••• | | | |
| VM202- 16 mg | XXXX | Date9. (Study Day) | Description | Yes/No |
| J | XXXX | Date9. (Study Day) | Description | Yes/No |

Note: Study Day = [(Date of Event) - (Treatment Start Date)]; 1 is added to the difference when 'Date of Event' is greater than or equal to 'Treatment Start Date'. path\t\_program.sas date time

Programmer note cause of death description includes AE#, for SAE, and specification for Other.